CLINICAL TRIAL: NCT03970733
Title: ALTERNATIVE SCHEDULE STUDY FOR VLA15, A MULTIVALENT RECOMBINANT OSPA BASED VACCINE CANDIDATE AGAINST LYME BORRELIOSIS, IN HEALTHY ADULTS AGED 18 TO 65 YEARS - A RANDOMIZED, CONTROLLED, OBSERVER-BLIND PHASE 2 STUDY.
Brief Title: Alternative Schedule Study For VLA15, a Vaccine Candidate Against Lyme Borreliosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA15-202; C4601007 (Other: Alias Study Number)
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Lyme Borreliosis
Keywords: VLA15; Lyme Borreliosis; Vaccine
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VLA15 with Alum lower dose (Experimental): Main Study Phase: VLA15 with Alum lower dose - Booster Phase: arm discontinued
  Interventions: Biological: VLA15
- VLA15 with Alum higher dose (Experimental): Main Study Phase: VLA15 with Alum higher dose - Booster Phase: VLA15 higher dose or placebo
  Interventions: Biological: VLA15
- Placebo (Placebo Comparator): Main Study Phase: placebo - Booster Phase: arm discontinued
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA15 — a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate
  Arms: VLA15 with Alum higher dose; VLA15 with Alum lower dose
Biological: Placebo — PBS (Phosphate Buffered Saline)
  Arms: Placebo

SUMMARY:
In the Main Study Phase a total of 246 subjects were randomized 2:2:1 into three treatment groups to receive either VLA15 with Alum (lower or higher dose) or Placebo. Main Study Phase vaccinations were administered as intramuscular injections on Day 1, Day 57 and Day 180.

In the Booster Phase subjects from the higher dose group who completed their primary immunization schedule according to protocol will be randomized 2:1 to receive an additional higher dose VLA15 vaccination or Placebo at Month 18.

Study duration in the Main Study Phase per subject is a maximum of 20 months. Overall study Duration is estimated to be 22 months.

Study duration per subject in the Booster Phase is a maximum of approximately 13 months.

Study duration per subject in the Main Study Phase and Booster Phase together is estimated to be a maximum of approximately 33 months.

Overall study duration (i.e., First-Subject-In to Last-Subject Out/ end of Booster Phase) is estimated to be approximately 37 months.

DETAILED DESCRIPTION:
This is a randomized, observer-blind (subject, Sponsor and investigator/site staff involved in Clinical Evaluation of subjects are blinded), Placebo controlled, multicenter Phase 2 study.

In Main Study Phase a total of 246 healthy subjects,aged 18 to 65 years, were randomized 2:2:1 to receive either VLA15 with Alum (lower or higher doser Placebo. Main Study Phase vaccinations were administered as intramuscular injections on Day 1 (Month 0), Day 57 (Month 2) and Day 180 (Month 6).

Subjects from the higher dose group who completed their primary immunization schedule according to protocol, will be randomized 2:1 to receive an additional injection of the higher dose VLA15 with Alum or Placebo in a Booster Phase. The additional vaccination is administered as intramuscular injection approximately 18 months after the first immunization.

ELIGIBILITY:
Inclusion Criteria - Main Study Phase:

* Subject is aged 18 to 65 years at the day of screening
* Subject is of good general health, including subjects with pharmacologically controlled chronic conditions;
* Subject has an understanding of the study and its procedures, agrees to its provisions,and gives written informed consent prior to any study-related procedures;
* If subject is of childbearing potential:
* Subject has a negative serum pregnancy test at screening;
* Subject agrees to employ adequate birth control measures for the duration of the study.

Inclusion Criteria - Booster Phase:

1. Randomization into higher dose group in the Main Study Phase
2. No relevant protocol deviation in the Main Study Phase, i.e., included in the Per-Protocol population for the Day 208 interim analysis of the Main Study;
3. Subject is of good general health, including subjects with pharmacologically controlled chronic conditions;
4. Subject has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures;
5. If subject is of childbearing potential:

   1. Subject has a negative Urine pregnancy test before booster vaccination;
   2. Subject agrees to employ adequate birth control measures for the duration of the study

Exclusion Criteria - Main Study Phase:

* Subject has a chronic illness related to Lyme borreliosis (LB), an active symptomatic LB as suspected or diagnosed by a physician, or received treatment for LB within the last 3 months prior to screening;
* Subject received previous vaccination against LB.;
* Subject had a tick bite within 4 weeks prior to vaccination visit;
* Subject has a medical history of or currently has a clinically relevant disease (e.g. cardiovascular, respiratory, neurologic, psychiatric conditions) which poses a risk for participation in the study, based on investigators judgement, such as individuals with poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment. Subjects with pharmacologically controlled conditions like osteoarthritis, depression, or asthma are eligible;
* Subject has a medical history of or currently has a neuroinflammatory or autoimmune disease, including Guillain Barré Syndrome;
* Subject has a known thrombocytopenia, bleeding disorder, or received anticoagulants in the three weeks prior to each study vaccination, contraindicating I.M. vaccination as judged by the investigator;
* Subject has received an active or passive immunization within 28 days before or after any vaccination; except for influenza (seasonal or pandemic) vaccines which may be administered outside a 7-days interval before or after any trial vaccination;
* Subject has received any other non-registered medicinal product in another clinical Trial within 28 days prior to VLA15 vaccination and throughout the entire study period or has received a registered medicinal product in another clinical Trial within 28 days prior to VLA15 vaccination and up to Day 208;
* Subject has a known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired immunodeficiency, including infection with human immunodeficiency virus (HIV), Status post organ transplantation or immuno-suppressive therapy within 30 days prior to first vaccination. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent >=0.05 mg/kg/day. Topical and inhaled steroids are allowed;
* Subject has a history of anaphylaxis or severe allergic reactions or a known hypersensitivity or allergic reactions to one of the components of the vaccine; Subject had any malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled;
* Subject had acute febrile infections within 10 days prior to first vaccination;
* Subject is pregnant (positive serum pregnancy test at screening), has plans to become pregnant during the course of the study or is lactating at the time of enrollment. Women of childbearing potential that are unwilling or unable to employ an adequate birth Control measure for the duration of the study.
* Subject has donated blood or blood-derived products (e.g. plasma) within 30 days or received blood or blood-derived products (e.g. plasma) within 90 days prior to first vaccination in this study or plans to donate or use blood or blood products during the course of the study;
* Subject has any condition that, in the opinion of the investigator, may compromise the subject's well-being, might interfere with evaluation of study endpoints, or would Limit the subject's ability to complete the study;
* Subject is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
* Subject is in a dependent relationship with the sponsor, an investigator or other study team member, or the study center. Dependent relationships include close relatives and household members (i.e. children, partner/spouse, siblings, parents) as well as employees of the investigator or study center personnel.

Exclusion Criteria - Booster Phase:

1. Subject met an individual stopping criterion during the Main Study Phase;
2. Subject has developed a chronic illness related to Lyme borreliosis (LB), an active symptomatic LB as suspected or diagnosed by a physician, or received treatment for LB within the last 3 months prior to vaccination visit;
3. Subject has developed a clinically relevant disease (e.g. cardiovascular, respiratory, neurologic, psychiatric conditions) which poses a risk for further participation in the study, based on investigators judgement, such as individuals with poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment;
4. Subject has developed a neuroinflammatory or autoimmune disease, including Guillain Barré Syndrome;
5. Subject has developed an immunodeficiency, including known infection with human immunodeficiency virus (HIV), status post organ transplantation, or immuno-suppressive therapy within 30 days prior to vaccination visit. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent >= 0.05 mg/kg/day. Topical and inhaled steroids are allowed;
6. Subject has developed anaphylaxis or severe allergic reactions;
7. Subject has developed allergic reactions to one of the components of the vaccine;
8. Subject has developed a malignancy;
9. Subject has developed thrombocytopenia or received anticoagulants in the 3 weeks prior to the booster vaccination contraindicating I.M. vaccination as judged by the investigator;
10. Subject has received any other non-registered medicinal product in another clinical trial within 28 days prior to VLA15 booster vaccination at Month 18 or plans to participate in another clinical trial with a non-registered medicinal product until Month 24;
11. Subject is pregnant, or plans to become pregnant prior to Month 24, or is lactating. Women of childbearing potential that are unwilling or unable to employ an adequate birth control measure for the duration of the study;
12. Subject has developed any condition that, in the opinion of the investigator, may compromise the subject's well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
13. Subject has been committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
14. Subject is in a dependent relationship with the sponsor, an investigator or other study team member, or the study center. Dependent relationships include close relatives and household members (i.e. children, partner/spouse, sibling).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc, Endwell, New York
  - Rochester Clinical Research, Inc., Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ghadge SK, Schneider M, Dubischar K, Wagner L, Kadlecek V, Obersriebnig M, Hochreiter R, Klingler A, Larcher-Senn J, Derhaschnig U, Bender W, Eder-Lingelbach S, Bezay N. Immunogenicity and safety of an 18-month booster dose of the VLA15 Lyme borreliosis vaccine candidate after primary immunisation in healthy adults in the USA: results of the booster phase of a randomised, controlled, phase 2 trial. Lancet Infect Dis. 2024 Nov;24(11):1275-1286. doi: 10.1016/S1473-3099(24)00372-4. Epub 2024 Jul 16. PMID 39029481
- [Derived] Bezay N, Wagner L, Kadlecek V, Obersriebnig M, Wressnigg N, Hochreiter R, Schneider M, Dubischar K, Derhaschnig U, Klingler A, Larcher-Senn J, Eder-Lingelbach S, Bender W. Optimisation of dose level and vaccination schedule for the VLA15 Lyme borreliosis vaccine candidate among healthy adults: two randomised, observer-blind, placebo-controlled, multicentre, phase 2 studies. Lancet Infect Dis. 2024 Sep;24(9):1045-1058. doi: 10.1016/S1473-3099(24)00175-0. Epub 2024 May 31. PMID 38830375
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=VLA15-202

RESULTS

PARTICIPANT FLOW:
Groups:
- VLA15 With Alum Lower Dose: Main Study Phase: VLA15 with Alum lower dose - Booster Phase: arm discontinued VLA15: a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate.
- VLA15 With Alum Higher Dose: Main Study Phase: VLA15 with Alum higher dose - Booster Phase: VLA15 higher dose or placebo VLA15: a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate.
- Placebo: Main Study Phase: placebo - Booster phase: arm discontinued Placebo: PBS (Phosphate Buffered Saline).
- Booster Phase: VLA15 With Alum Higher Dose: Participants who received higher dose of VLA15 with alum in main study phase were randomized to receive a single booster dose of VLA15 with alum higher dose vaccine at Month 18 in booster phase.
- Booster Phase: Placebo: Participants who received higher dose of VLA15 with alum in main study phase were randomized to receive a single dose of placebo at Month 18 in booster phase.
Period: Main Study Phase (18 Months)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Started | 97 | 98 | 51 | 0 | 0
Completed (Participants who completed Day 545 (Month 18)) | 89 | 84 | 46 | 0 (No participants were enrolled in this arm during the main study phase.) | 0 (No participants were enrolled in this arm during the main study phase.)
Not Completed | 8 | 14 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 2 | 0 | 0
Not completed — Moved from study area | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 5 | 3 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0
Period: Booster Phase (Approx. 12 Months)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Started | 0 (Participants did not continue booster phase.) | 0 (Participants who continued to booster phase are reported under booster phase arms.) | 0 (Participants did not continue booster phase.) | 39 | 19
Completed | 0 | 0 | 0 | 39 | 18
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Groups:
- VLA15 With Alum Lower Dose: 0.75 ml injection of VLA15 w/ alum applied at Days 1, 57, and 180 in the Main study phase. VLA15 is a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate. Participants of this arm did not enter booster phase.
- VLA15 With Alum Higher Dose: 1 ml injection of VLA15 w/ alum applied at Days 1, 57, and 180 in the Main study phase. VLA15 is a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate. Participants after completing main study, upon consent were randomized to receive either VLA15 with Alum higher dose arm or Placebo in booster phase.
- Placebo: 1 ml injection of placebo applied at Days 1, 57, and 180 in the Main study phase. Placebo: phosphate buffered saline (PBS) solution. Participants of this arm did not enter booster phase.
- Total: Total of all reporting groups
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo | Total
Number analyzed (Participants) | 97 | 98 | 51 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Here, number analyzed signifies number of participants evaluable for specified rows.
  years
    Main Study Phase | 43.5 (12.61) | 43.0 (12.76) | 45.0 (12.79) | 43.6 (12.68)
    Booster Phase: VLA15 with Alum higher dose: number analyzed (Participants) | 0 | 39 | 0 | 39
    Booster Phase: VLA15 with Alum higher dose |  | 46.5 (13.15) |  | 46.5 (13.15)
    Booster Phase: Placebo: number analyzed (Participants) | 0 | 19 | 0 | 19
    Booster Phase: Placebo |  | 38.8 (13.50) |  | 38.8 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows.
  Participants
    Main Study Phase: Female | 49 | 50 | 34 | 133
    Main Study Phase: Male | 48 | 48 | 17 | 113
    Booster Phase: VLA15 with Alum higher dose: number analyzed (Participants) | 0 | 39 | 0 | 39
    Booster Phase: VLA15 with Alum higher dose: Female | 0 | 23 | 0 | 23
    Booster Phase: VLA15 with Alum higher dose: Male | 0 | 16 | 0 | 16
    Booster Phase: Placebo: number analyzed (Participants) | 0 | 19 | 0 | 19
    Booster Phase: Placebo: Female | 0 | 7 | 0 | 7
    Booster Phase: Placebo: Male | 0 | 12 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows.
  Participants
    Main Study Phase: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Main Study Phase: Asian | 0 | 1 | 0 | 1
    Main Study Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Main Study Phase: Black or African American | 4 | 4 | 0 | 8
    Main Study Phase: White | 91 | 93 | 51 | 235
    Main Study Phase: More than one race | 0 | 0 | 0 | 0
    Main Study Phase: Unknown or Not Reported | 2 | 0 | 0 | 2
    Booster Phase: VLA15 with Alum higher dose: number analyzed (Participants) | 0 | 39 | 0 | 39
    Booster Phase: VLA15 with Alum higher dose: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Booster Phase: VLA15 with Alum higher dose: Asian | 0 | 1 | 0 | 1
    Booster Phase: VLA15 with Alum higher dose: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Booster Phase: VLA15 with Alum higher dose: Black or African American | 0 | 4 | 0 | 4
    Booster Phase: VLA15 with Alum higher dose: White | 0 | 34 | 0 | 34
    Booster Phase: VLA15 with Alum higher dose: More than one race | 0 | 0 | 0 | 0
    Booster Phase: VLA15 with Alum higher dose: Unknown or Not Reported | 0 | 0 | 0 | 0
    Booster Phase: Placebo: number analyzed (Participants) | 0 | 19 | 0 | 19
    Booster Phase: Placebo: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Booster Phase: Placebo: Asian | 0 | 0 | 0 | 0
    Booster Phase: Placebo: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Booster Phase: Placebo: Black or African American | 0 | 0 | 0 | 0
    Booster Phase: Placebo: White | 0 | 19 | 0 | 19
    Booster Phase: Placebo: More than one race | 0 | 0 | 0 | 0
    Booster Phase: Placebo: Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: GMTs for IgG Against Each OspA Serotype
Description: Geometric Mean Titers (GMTs) for Immunoglobulin G (IgG) against each Outer Surface Protein A (OspA) serotype ST1 to ST6, determined by Enzyme-Linked Immunosorbent Assay (ELISA) at Day 208 (Month 7)
Time Frame: Day 208 (Month 7)
Population: Per-protocol population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 78 | 80 | 38
Units per milliliter (U/mL)
  ST1 Day 208 | 278.5 [214.9 to 361.0] | 274.7 [209.4 to 360.4] | 21.0 [19.6 to 22.5]
  ST2 Day 208 | 545.2 [431.8 to 688.4] | 579.8 [461.9 to 727.8] | 20.0 [20.0 to 20.0]
  ST3 Day 208 | 520.0 [410.5 to 658.7] | 596.8 [471.9 to 754.8] | 20.0 [20.0 to 20.0]
  ST4 Day 208 | 332.6 [261.3 to 423.3] | 367.8 [293.8 to 460.4] | 21.3 [19.8 to 23.0]
  ST5 Day 208 | 332.8 [262.9 to 421.3] | 358.8 [283.7 to 453.7] | 20.0 [20.0 to 20.0]
  ST6 Day 208 | 339.9 [267.3 to 432.3] | 345.7 [273.7 to 436.6] | 21.4 [19.4 to 23.5]

2. Secondary Outcome: GMTs for IgG Against Each OspA Serotype During the Main Study Phase
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 365 (Month 12) and 545 (Month 18).
Time Frame: At Day 1 (Month 0), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 365 (Month 12) and Day 545 (Month 18)
Population: Per-protocol population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity). Here, "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 85 | 86 | 43
Units per milliliter (U/mL)
  ST1 Day 1 | 21.4 [19.8 to 23.1] | 20.2 [19.8 to 20.6] | 21.8 [19.6 to 24.1]
  ST1 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST1 Day 29 | 22.0 [20.2 to 24.0] | 20.4 [19.8 to 21.0] | 22.1 [19.9 to 24.6]
  ST1 Day 57 | 22.5 [20.6 to 24.6] | 21.1 [19.9 to 22.3] | 21.6 [19.6 to 23.9]
  ST1 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST1 Day 85 | 64.5 [50.7 to 82.0] | 75.2 [59.6 to 94.9] | 21.7 [19.7 to 23.8]
  ST1 Day 180 | 26.4 [23.0 to 30.2] | 24.9 [22.7 to 27.4] | 21.5 [19.7 to 23.4]
  ST1 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST1 Day 365 | 48.3 [39.1 to 59.7] | 37.2 [30.6 to 45.2] | 21.4 [19.8 to 23.1]
  ST1 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST1 Day 545 | 29.7 [24.4 to 36.3] | 23.9 [21.5 to 26.7] | 20.6 [19.4 to 21.9]
  ST2 Day 1 | 20.8 [19.9 to 21.8] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST2 Day 29 | 21.5 [20.2 to 23.0] | 21.9 [20.2 to 23.6] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 21.3 [20.0 to 22.6] | 22.0 [20.1 to 24.0] | 20.0 [20.0 to 20.0]
  ST2 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST2 Day 85 | 162.6 [127.0 to 208.2] | 183.5 [144.9 to 232.4] | 20.0 [20.0 to 20.0]
  ST2 Day 180 | 38.0 [30.9 to 46.5] | 35.4 [29.9 to 41.9] | 20.0 [20.0 to 20.0]
  ST2 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST2 Day 365 | 87.2 [69.0 to 110.2] | 71.1 [57.0 to 88.8] | 20.0 [20.0 to 20.0]
  ST2 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST2 Day 545 | 44.6 [35.9 to 55.4] | 33.1 [27.5 to 39.7] | 21.1 [19.0 to 23.4]
  ST3 Day 1 | 20.3 [19.8 to 20.8] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST3 Day 29 | 21.3 [20.0 to 22.7] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 20.9 [19.8 to 22.1] | 20.7 [19.3 to 22.3] | 20.0 [20.0 to 20.0]
  ST3 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST3 Day 85 | 166.3 [128.6 to 215.0] | 217.7 [171.7 to 275.9] | 20.7 [19.3 to 22.2]
  ST3 Day 180 | 38.2 [31.6 to 46.1] | 41.0 [34.7 to 48.5] | 20.4 [19.6 to 21.4]
  ST3 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST3 Day 365 | 78.5 [62.7 to 98.3] | 74.6 [59.6 to 93.3] | 20.0 [20.0 to 20.0]
  ST3 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST3 Day 545 | 39.1 [31.9 to 48.0] | 32.2 [27.4 to 37.8] | 20.0 [20.0 to 20.0]
  ST4 Day 1 | 20.7 [19.7 to 21.7] | 20.3 [19.7 to 21.0] | 20.5 [19.5 to 21.7]
  ST4 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST4 Day 29 | 20.8 [19.7 to 21.9] | 20.5 [19.8 to 21.3] | 20.8 [19.7 to 22.0]
  ST4 Day 57 | 21.0 [20.0 to 22.1] | 20.9 [19.8 to 22.1] | 21.2 [19.8 to 22.8]
  ST4 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST4 Day 85 | 79.3 [63.2 to 99.6] | 100.8 [81.2 to 125.0] | 21.6 [20.0 to 23.3]
  ST4 Day 180 | 28.0 [24.6 to 31.9] | 27.1 [24.1 to 30.4] | 21.3 [19.8 to 22.8]
  ST4 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST4 Day 365 | 53.9 [44.1 to 65.9] | 43.2 [35.5 to 52.5] | 21.0 [19.6 to 22.5]
  ST4 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST4 Day 545 | 35.5 [29.7 to 42.5] | 27.3 [24.0 to 31.1] | 22.4 [19.3 to 26.1]
  ST5 Day 1 | 21.0 [19.9 to 22.2] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST5 Day 29 | 21.5 [20.0 to 23.1] | 20.9 [19.8 to 22.0] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 21.3 [20.0 to 22.7] | 21.3 [19.9 to 22.9] | 20.0 [20.0 to 20.0]
  ST5 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST5 Day 85 | 87.4 [69.1 to 110.5] | 100.2 [81.0 to 124.1] | 20.0 [20.0 to 20.0]
  ST5 Day 180 | 29.0 [24.9 to 33.8] | 27.0 [24.1 to 30.3] | 20.0 [20.0 to 20.0]
  ST5 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST5 Day 365 | 53.9 [43.5 to 66.9] | 42.7 [34.9 to 52.2] | 20.0 [20.0 to 20.0]
  ST5 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST5 Day 545 | 35.0 [28.9 to 42.4] | 27.1 [23.8 to 30.9] | 20.4 [19.6 to 21.2]
  ST6 Day 1 | 22.6 [20.6 to 24.8] | 20.7 [19.7 to 21.6] | 21.2 [19.5 to 23.1]
  ST6 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST6 Day 29 | 23.3 [20.9 to 25.9] | 21.2 [20.0 to 22.4] | 21.0 [19.6 to 22.5]
  ST6 Day 57 | 23.2 [21.0 to 25.6] | 22.2 [20.5 to 24.2] | 21.6 [19.8 to 23.6]
  ST6 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST6 Day 85 | 79.9 [62.9 to 101.5] | 84.3 [67.4 to 105.4] | 20.7 [19.3 to 22.1]
  ST6 Day 180 | 32.7 [27.8 to 38.4] | 28.8 [25.3 to 32.7] | 21.7 [19.7 to 23.9]
  ST6 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST6 Day 365 | 61.1 [48.9 to 76.3] | 46.7 [37.9 to 57.5] | 21.5 [19.8 to 23.4]
  ST6 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST6 Day 545 | 36.8 [30.0 to 45.3] | 27.1 [23.6 to 31.1] | 20.7 [19.3 to 22.1]

3. Secondary Outcome: SCRs for Each OspA Serotype Specific IgG During the Main Study Phase
Description: Seroconversion Rate (SCR) for each Outer Surface Protein A (OspA) serotype specific IgG ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18). Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): greater than or equal to (>=) 4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants. Percentages are based on the number of participants with non-missing observations.
Time Frame: Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12) and Day 545 (Month 18)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 85 | 86 | 43
Percentage of Participants
  ST1 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST1 Day 29 | 2.4 [0.7 to 8.4] | 1.2 [0.2 to 6.3] | 2.3 [0.4 to 12.1]
  ST1 Day 57 | 4.7 [1.8 to 11.5] | 3.5 [1.2 to 9.8] | 0.0 [0.0 to 8.2]
  ST1 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST1 Day 85 | 59.0 [48.3 to 69.0] | 69.0 [58.5 to 77.9] | 2.3 [0.4 to 12.1]
  ST1 Day 180 | 14.1 [8.3 to 23.1] | 19.8 [12.7 to 29.4] | 4.7 [1.3 to 15.5]
  ST1 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST1 Day 208 | 92.3 [84.2 to 96.4] | 93.8 [86.2 to 97.3] | 0.0 [0.0 to 9.2]
  ST1 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST1 Day 365 | 50.0 [39.4 to 60.6] | 38.0 [28.1 to 49.0] | 2.4 [0.4 to 12.3]
  ST1 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST1 Day 545 | 17.8 [10.7 to 28.1] | 13.8 [7.5 to 24.3] | 0.0 [0.0 to 9.2]
  ST2 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST2 Day 29 | 2.4 [0.7 to 8.4] | 5.8 [2.5 to 12.9] | 0.0 [0.0 to 8.2]
  ST2 Day 57 | 1.2 [0.2 to 6.4] | 5.8 [2.5 to 12.9] | 0.0 [0.0 to 8.2]
  ST2 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST2 Day 85 | 84.3 [75.0 to 90.6] | 89.3 [80.9 to 94.3] | 0.0 [0.0 to 8.2]
  ST2 Day 180 | 32.9 [23.9 to 43.5] | 38.4 [28.8 to 48.9] | 0.0 [0.0 to 8.2]
  ST2 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST2 Day 208 | 96.2 [89.3 to 98.7] | 98.8 [93.3 to 99.8] | 0.0 [0.0 to 9.2]
  ST2 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST2 Day 365 | 72.0 [61.4 to 80.5] | 70.9 [60.1 to 79.7] | 0.0 [0.0 to 8.4]
  ST2 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST2 Day 545 | 45.2 [34.3 to 56.6] | 35.4 [24.9 to 47.5] | 2.6 [0.5 to 13.5]
  ST3 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST3 Day 29 | 3.6 [1.2 to 10.1] | 0.0 [0.0 to 4.3] | 0.0 [0.0 to 8.2]
  ST3 Day 57 | 2.4 [0.6 to 8.2] | 1.2 [0.2 to 6.3] | 0.0 [0.0 to 8.2]
  ST3 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST3 Day 85 | 84.3 [75.0 to 90.6] | 91.7 [83.8 to 95.9] | 2.3 [0.4 to 12.1]
  ST3 Day 180 | 40.0 [30.2 to 50.6] | 50.0 [39.7 to 60.3] | 2.3 [0.4 to 12.1]
  ST3 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST3 Day 208 | 98.7 [93.1 to 99.8] | 97.5 [91.3 to 99.3] | 0.0 [0.0 to 9.2]
  ST3 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST3 Day 365 | 70.7 [60.1 to 79.5] | 70.9 [60.1 to 79.7] | 0.0 [0.0 to 8.4]
  ST3 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST3 Day 545 | 42.5 [31.8 to 53.9] | 36.9 [26.2 to 49.1] | 0.0 [0.0 to 9.2]
  ST4 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST4 Day 29 | 1.2 [0.2 to 6.5] | 1.2 [0.2 to 6.3] | 2.3 [0.4 to 12.1]
  ST4 Day 57 | 2.4 [0.6 to 8.2] | 2.3 [0.6 to 8.1] | 4.7 [1.3 to 15.5]
  ST4 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST4 Day 85 | 74.7 [64.4 to 82.8] | 83.3 [73.9 to 89.8] | 7.0 [2.4 to 18.6]
  ST4 Day 180 | 25.9 [17.8 to 36.1] | 24.4 [16.6 to 34.5] | 4.7 [1.3 to 15.5]
  ST4 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST4 Day 208 | 97.4 [91.1 to 99.3] | 98.8 [93.3 to 99.8] | 5.3 [1.5 to 17.3]
  ST4 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST4 Day 365 | 62.2 [51.4 to 71.9] | 51.9 [41.1 to 62.6] | 2.4 [0.4 to 12.3]
  ST4 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST4 Day 545 | 39.7 [29.3 to 51.2] | 27.7 [18.3 to 39.6] | 5.3 [1.5 to 17.3]
  ST5 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST5 Day 29 | 1.2 [0.2 to 6.5] | 3.5 [1.2 to 9.8] | 0.0 [0.0 to 8.2]
  ST5 Day 57 | 1.2 [0.2 to 6.4] | 4.7 [1.8 to 11.4] | 0.0 [0.0 to 8.2]
  ST5 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST5 Day 85 | 73.5 [63.1 to 81.8] | 81.0 [71.3 to 87.9] | 0.0 [0.0 to 8.2]
  ST5 Day 180 | 20.0 [12.9 to 29.7] | 25.6 [17.5 to 35.7] | 0.0 [0.0 to 8.2]
  ST5 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST5 Day 208 | 94.9 [87.5 to 98.0] | 96.3 [89.5 to 98.7] | 0.0 [0.0 to 9.2]
  ST5 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST5 Day 365 | 53.7 [42.9 to 64.0] | 48.1 [37.4 to 58.9] | 0.0 [0.0 to 8.4]
  ST5 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST5 Day 545 | 34.2 [24.4 to 45.7] | 27.7 [18.3 to 39.6] | 2.6 [0.5 to 13.5]
  ST6 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST6 Day 29 | 2.4 [0.7 to 8.4] | 2.3 [0.6 to 8.1] | 2.3 [0.4 to 12.1]
  ST6 Day 57 | 3.5 [1.2 to 9.9] | 5.8 [2.5 to 12.9] | 4.7 [1.3 to 15.5]
  ST6 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST6 Day 85 | 61.4 [50.7 to 71.2] | 71.4 [61.0 to 80.0] | 0.0 [0.0 to 8.2]
  ST6 Day 180 | 27.1 [18.8 to 37.3] | 26.7 [18.5 to 36.9] | 4.7 [1.3 to 15.5]
  ST6 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST6 Day 208 | 89.7 [81.0 to 94.7] | 96.3 [89.5 to 98.7] | 2.6 [0.5 to 13.5]
  ST6 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST6 Day 365 | 56.1 [45.3 to 66.3] | 49.4 [38.6 to 60.2] | 4.8 [1.3 to 15.8]
  ST6 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST6 Day 545 | 31.5 [22.0 to 42.9] | 21.5 [13.3 to 33.0] | 0.0 [0.0 to 9.2]

4. Secondary Outcome: GMFR as Compared to Baseline for IgG Against Each OspA Serotype During the Main Study Phase
Description: Geometric Mean Fold Rise (GMFR) as compared to baseline for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18).
Time Frame: Day 1 (baseline from where comparison was done), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12) and Day 545 (Month 18)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 85 | 86 | 43
Fold Rise
  ST1 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST1 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1]
  ST1 Day 57 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST1 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST1 Day 85 | 3.0 [2.4 to 3.8] | 3.7 [3.0 to 4.7] | 1.0 [0.9 to 1.1]
  ST1 Day 180 | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 1.0 [0.9 to 1.1]
  ST1 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST1 Day 208 | 12.9 [9.8 to 17.1] | 13.6 [10.4 to 17.8] | 1.0 [0.9 to 1.0]
  ST1 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST1 Day 365 | 2.3 [1.8 to 2.8] | 1.8 [1.5 to 2.2] | 1.0 [0.9 to 1.1]
  ST1 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST1 Day 545 | 1.4 [1.1 to 1.7] | 1.2 [1.1 to 1.3] | 0.9 [0.9 to 1.0]
  ST2 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST2 Day 29 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST2 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST2 Day 85 | 7.8 [6.1 to 10.0] | 9.2 [7.2 to 11.6] | 1.0 [1.0 to 1.0]
  ST2 Day 180 | 1.8 [1.5 to 2.2] | 1.8 [1.5 to 2.1] | 1.0 [1.0 to 1.0]
  ST2 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST2 Day 208 | 26.1 [20.4 to 33.3] | 29.0 [23.1 to 36.4] | 1.0 [1.0 to 1.0]
  ST2 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST2 Day 365 | 4.2 [3.3 to 5.3] | 3.6 [2.8 to 4.4] | 1.0 [1.0 to 1.0]
  ST2 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST2 Day 545 | 2.1 [1.7 to 2.6] | 1.7 [1.4 to 2.0] | 1.1 [0.9 to 1.2]
  ST3 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST3 Day 29 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST3 Day 57 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST3 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST3 Day 85 | 8.2 [6.3 to 10.6] | 10.9 [8.6 to 13.8] | 1.0 [1.0 to 1.1]
  ST3 Day 180 | 1.9 [1.6 to 2.3] | 2.1 [1.7 to 2.4] | 1.0 [1.0 to 1.1]
  ST3 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST3 Day 208 | 25.6 [20.2 to 32.6] | 29.8 [23.6 to 37.7] | 1.0 [1.0 to 1.0]
  ST3 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST3 Day 365 | 3.9 [3.1 to 4.9] | 3.7 [3.0 to 4.7] | 1.0 [1.0 to 1.0]
  ST3 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST3 Day 545 | 2.0 [1.6 to 2.4] | 1.6 [1.4 to 1.9] | 1.0 [1.0 to 1.0]
  ST4 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST4 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST4 Day 57 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1]
  ST4 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST4 Day 85 | 3.8 [3.1 to 4.8] | 5.0 [4.0 to 6.1] | 1.1 [1.0 to 1.1]
  ST4 Day 180 | 1.4 [1.2 to 1.5] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.1]
  ST4 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST4 Day 208 | 16.0 [12.6 to 20.4] | 18.1 [14.5 to 22.6] | 1.0 [1.0 to 1.1]
  ST4 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST4 Day 365 | 2.6 [2.1 to 3.2] | 2.1 [1.8 to 2.6] | 1.0 [1.0 to 1.1]
  ST4 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST4 Day 545 | 1.7 [1.4 to 2.0] | 1.3 [1.2 to 1.5] | 1.1 [0.9 to 1.3]
  ST5 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST5 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST5 Day 85 | 4.2 [3.3 to 5.2] | 5.0 [4.0 to 6.2] | 1.0 [1.0 to 1.0]
  ST5 Day 180 | 1.4 [1.2 to 1.6] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.0]
  ST5 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST5 Day 208 | 15.8 [12.4 to 20.0] | 17.9 [14.2 to 22.7] | 1.0 [1.0 to 1.0]
  ST5 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST5 Day 365 | 2.6 [2.1 to 3.2] | 2.1 [1.7 to 2.6] | 1.0 [1.0 to 1.0]
  ST5 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST5 Day 545 | 1.7 [1.4 to 2.0] | 1.4 [1.2 to 1.5] | 1.0 [1.0 to 1.1]
  ST6 Day 29: number analyzed (Participants) | 83 | 86 | 43
  ST6 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [0.9 to 1.1]
  ST6 Day 57 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.2] | 1.0 [0.9 to 1.1]
  ST6 Day 85: number analyzed (Participants) | 83 | 84 | 43
  ST6 Day 85 | 3.5 [2.8 to 4.5] | 4.1 [3.3 to 5.1] | 1.0 [0.9 to 1.0]
  ST6 Day 180 | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.6] | 1.0 [0.9 to 1.1]
  ST6 Day 208: number analyzed (Participants) | 78 | 80 | 38
  ST6 Day 208 | 14.9 [11.4 to 19.3] | 16.7 [13.2 to 21.1] | 1.0 [0.9 to 1.1]
  ST6 Day 365: number analyzed (Participants) | 82 | 79 | 42
  ST6 Day 365 | 2.7 [2.1 to 3.4] | 2.3 [1.8 to 2.8] | 1.0 [0.9 to 1.1]
  ST6 Day 545: number analyzed (Participants) | 73 | 65 | 38
  ST6 Day 545 | 1.6 [1.3 to 1.9] | 1.3 [1.1 to 1.5] | 1.0 [0.9 to 1.0]

5. Secondary Outcome: GMTs for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 18 - 49 Years
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 18 - 49 years.
Time Frame: At Day 1 (Month 0), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12) and Day 545 (Month 18)
Population: Per-protocol population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 55 | 57 | 30
Units per milliliter (U/mL)
  ST1 Day 1 | 20.8 [19.3 to 22.4] | 20.3 [19.7 to 20.9] | 21.2 [19.5 to 23.1]
  ST1 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST1 Day 29 | 21.3 [19.5 to 23.4] | 20.6 [19.8 to 21.5] | 21.2 [19.5 to 23.1]
  ST1 Day 57 | 22.0 [19.9 to 24.3] | 20.9 [19.9 to 22.0] | 21.0 [19.6 to 22.5]
  ST1 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST1 Day 85 | 60.8 [43.6 to 84.8] | 83.6 [61.7 to 113.2] | 21.3 [19.5 to 23.2]
  ST1 Day 180 | 27.2 [22.7 to 32.5] | 25.1 [22.2 to 28.4] | 21.0 [19.6 to 22.6]
  ST1 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST1 Day 208 | 284.1 [203.4 to 396.9] | 291.2 [211.6 to 400.8] | 20.6 [19.4 to 21.9]
  ST1 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST1 Day 365 | 47.8 [36.4 to 62.7] | 37.4 [29.7 to 47.1] | 21.2 [19.5 to 23.1]
  ST1 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST1 Day 545 | 30.9 [23.3 to 41.0] | 23.5 [20.6 to 26.6] | 20.0 [20.0 to 20.0]
  ST2 Day 1 | 20.4 [19.6 to 21.3] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST2 Day 29 | 21.5 [19.8 to 23.3] | 21.7 [19.8 to 23.9] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 20.9 [19.6 to 22.3] | 22.5 [19.9 to 25.4] | 20.0 [20.0 to 20.0]
  ST2 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST2 Day 85 | 155.9 [113.0 to 215.0] | 195.1 [145.0 to 262.6] | 20.0 [20.0 to 20.0]
  ST2 Day 180 | 36.6 [28.9 to 46.4] | 36.0 [29.2 to 44.3] | 20.0 [20.0 to 20.0]
  ST2 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST2 Day 208 | 551.9 [419.0 to 727.0] | 581.3 [465.3 to 726.2] | 20.0 [20.0 to 20.0]
  ST2 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST2 Day 365 | 82.6 [62.2 to 109.7] | 66.1 [51.2 to 85.5] | 20.0 [20.0 to 20.0]
  ST2 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST2 Day 545 | 46.3 [35.3 to 60.8] | 32.3 [26.1 to 39.8] | 21.6 [18.5 to 25.2]
  ST3 Day 1 | 20.4 [19.6 to 21.2] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST3 Day 29 | 21.7 [19.7 to 23.8] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 21.1 [19.5 to 22.8] | 21.1 [18.9 to 23.6] | 20.0 [20.0 to 20.0]
  ST3 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST3 Day 85 | 178.3 [127.9 to 248.5] | 233.5 [172.9 to 315.2] | 21.0 [19.0 to 23.3]
  ST3 Day 180 | 40.3 [31.4 to 51.8] | 42.6 [34.5 to 52.6] | 20.6 [19.3 to 22.0]
  ST3 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST3 Day 208 | 573.5 [434.9 to 756.2] | 633.4 [507.5 to 790.6] | 20.0 [20.0 to 20.0]
  ST3 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST3 Day 365 | 80.2 [60.2 to 106.8] | 71.3 [54.7 to 92.9] | 20.0 [20.0 to 20.0]
  ST3 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST3 Day 545 | 40.8 [30.8 to 54.0] | 33.5 [27.1 to 41.3] | 20.0 [20.0 to 20.0]
  ST4 Day 1 | 21.0 [19.6 to 22.6] | 20.5 [19.5 to 21.5] | 20.8 [19.2 to 22.4]
  ST4 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST4 Day 29 | 21.2 [19.5 to 23.0] | 20.8 [19.7 to 21.9] | 20.7 [19.3 to 22.1]
  ST4 Day 57 | 21.3 [19.8 to 23.0] | 21.4 [19.7 to 23.2] | 21.8 [19.7 to 24.1]
  ST4 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST4 Day 85 | 84.4 [62.1 to 114.5] | 111.9 [85.1 to 147.2] | 21.7 [19.8 to 23.9]
  ST4 Day 180 | 29.3 [24.5 to 35.2] | 27.7 [23.8 to 32.2] | 21.8 [19.7 to 24.1]
  ST4 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST4 Day 208 | 365.2 [275.1 to 484.8] | 393.3 [311.9 to 495.8] | 22.0 [19.7 to 24.5]
  ST4 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST4 Day 365 | 55.4 [42.7 to 72.0] | 42.6 [33.9 to 53.4] | 21.5 [19.4 to 23.8]
  ST4 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST4 Day 545 | 40.9 [31.8 to 52.6] | 28.0 [23.7 to 33.0] | 23.6 [18.9 to 29.5]
  ST5 Day 1 | 21.1 [19.6 to 22.6] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST5 Day 29 | 21.9 [19.7 to 24.2] | 20.4 [19.6 to 21.1] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 21.5 [19.7 to 23.4] | 21.3 [19.3 to 23.5] | 20.0 [20.0 to 20.0]
  ST5 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST5 Day 85 | 91.0 [66.9 to 123.7] | 106.4 [81.0 to 139.6] | 20.0 [20.0 to 20.0]
  ST5 Day 180 | 30.0 [24.6 to 36.6] | 27.1 [23.5 to 31.3] | 20.0 [20.0 to 20.0]
  ST5 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST5 Day 208 | 358.8 [269.7 to 477.4] | 371.0 [287.6 to 478.4] | 20.0 [20.0 to 20.0]
  ST5 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST5 Day 365 | 54.5 [40.9 to 72.5] | 42.0 [33.3 to 53.1] | 20.0 [20.0 to 20.0]
  ST5 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST5 Day 545 | 37.7 [28.8 to 49.4] | 26.8 [22.8 to 31.6] | 20.6 [19.4 to 21.8]
  ST6 Day 1 | 23.0 [20.2 to 26.3] | 20.6 [19.5 to 21.7] | 21.0 [19.0 to 23.3]
  ST6 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST6 Day 29 | 24.1 [20.6 to 28.0] | 21.0 [19.6 to 22.5] | 20.9 [19.1 to 22.8]
  ST6 Day 57 | 23.5 [20.5 to 26.9] | 22.5 [20.1 to 25.3] | 21.6 [19.4 to 24.0]
  ST6 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST6 Day 85 | 86.8 [63.6 to 118.4] | 85.4 [64.0 to 114.1] | 21.0 [19.0 to 23.1]
  ST6 Day 180 | 32.9 [26.5 to 40.8] | 27.5 [23.5 to 32.1] | 21.6 [19.3 to 24.3]
  ST6 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST6 Day 208 | 362.4 [277.1 to 473.9] | 337.5 [258.2 to 441.1] | 21.2 [18.8 to 23.8]
  ST6 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST6 Day 365 | 61.2 [45.9 to 81.8] | 41.7 [32.7 to 53.2] | 21.6 [19.3 to 24.1]
  ST6 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST6 Day 545 | 41.1 [30.7 to 55.0] | 24.7 [21.2 to 28.9] | 21.0 [19.0 to 23.1]

6. Secondary Outcome: GMTs for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 50 - 65 Years
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 50 - 65 years.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 30 | 29 | 13
Units per milliliter (U/mL)
  ST1 Day 1 | 22.6 [19.0 to 26.8] | 20.0 [20.0 to 20.0] | 23.1 [16.9 to 31.5]
  ST1 Day 29 | 23.3 [19.6 to 27.8] | 20.0 [20.0 to 20.0] | 24.4 [17.7 to 33.8]
  ST1 Day 57 | 23.5 [19.5 to 28.3] | 21.4 [18.6 to 24.6] | 23.2 [16.8 to 31.9]
  ST1 Day 85 | 71.5 [51.2 to 100.0] | 61.6 [42.8 to 88.5] | 22.6 [17.3 to 29.6]
  ST1 Day 180 | 24.9 [20.1 to 30.9] | 24.5 [20.9 to 28.6] | 22.5 [17.4 to 29.1]
  ST1 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST1 Day 208 | 269.3 [174.1 to 416.5] | 246.6 [145.6 to 417.5] | 21.9 [18.0 to 26.6]
  ST1 Day 365 | 49.2 [34.4 to 70.4] | 36.8 [25.3 to 53.4] | 21.8 [18.1 to 26.2]
  ST1 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST1 Day 545 | 27.9 [21.4 to 36.5] | 24.8 [20.1 to 30.5] | 21.9 [17.9 to 26.9]
  ST2 Day 1 | 21.6 [19.3 to 24.2] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29 | 21.7 [19.3 to 24.4] | 22.1 [19.0 to 25.7] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 21.9 [19.2 to 25.0] | 21.1 [18.9 to 23.5] | 20.0 [20.0 to 20.0]
  ST2 Day 85 | 175.3 [117.0 to 262.6] | 163.4 [108.4 to 246.1] | 20.0 [20.0 to 20.0]
  ST2 Day 180 | 40.5 [27.2 to 60.4] | 34.3 [25.4 to 46.3] | 20.0 [20.0 to 20.0]
  ST2 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST2 Day 208 | 534.1 [342.5 to 832.8] | 577.0 [340.7 to 977.2] | 20.0 [20.0 to 20.0]
  ST2 Day 365 | 95.9 [62.4 to 147.5] | 80.6 [52.4 to 124.2] | 20.0 [20.0 to 20.0]
  ST2 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST2 Day 545 | 41.9 [28.5 to 61.7] | 34.5 [23.9 to 49.7] | 20.0 [20.0 to 20.0]
  ST3 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29 | 20.6 [19.4 to 21.9] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 20.6 [19.4 to 21.8] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 85 | 147.1 [96.3 to 224.7] | 190.6 [127.1 to 285.7] | 20.0 [20.0 to 20.0]
  ST3 Day 180 | 34.5 [25.8 to 46.2] | 38.1 [28.4 to 51.0] | 20.0 [20.0 to 20.0]
  ST3 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST3 Day 208 | 440.6 [281.3 to 690.1] | 534.3 [307.0 to 930.0] | 20.0 [20.0 to 20.0]
  ST3 Day 365 | 75.7 [51.5 to 111.2] | 80.6 [52.7 to 123.4] | 20.0 [20.0 to 20.0]
  ST3 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST3 Day 545 | 36.6 [27.0 to 49.7] | 30.1 [23.1 to 39.1] | 20.0 [20.0 to 20.0]
  ST4 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST4 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 21.1 [18.8 to 23.7]
  ST4 Day 57 | 20.5 [19.5 to 21.7] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST4 Day 85 | 71.1 [50.4 to 100.3] | 82.6 [57.9 to 117.7] | 21.3 [18.6 to 24.3]
  ST4 Day 180 | 25.7 [21.8 to 30.3] | 25.9 [21.6 to 31.0] | 20.0 [20.0 to 20.0]
  ST4 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST4 Day 208 | 283.9 [179.8 to 448.3] | 324.8 [197.4 to 534.3] | 20.0 [20.0 to 20.0]
  ST4 Day 365 | 51.4 [37.0 to 71.4] | 44.3 [30.2 to 64.8] | 20.0 [20.0 to 20.0]
  ST4 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST4 Day 545 | 28.3 [22.6 to 35.5] | 26.3 [21.2 to 32.7] | 20.0 [20.0 to 20.0]
  ST5 Day 1 | 20.9 [19.1 to 22.8] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29 | 20.8 [19.2 to 22.7] | 21.9 [19.0 to 25.3] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 20.9 [19.1 to 23.0] | 21.4 [19.4 to 23.7] | 20.0 [20.0 to 20.0]
  ST5 Day 85 | 81.4 [55.9 to 118.5] | 89.6 [62.6 to 128.2] | 20.0 [20.0 to 20.0]
  ST5 Day 180 | 27.3 [21.3 to 34.9] | 26.7 [21.8 to 32.8] | 20.0 [20.0 to 20.0]
  ST5 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST5 Day 208 | 293.1 [190.5 to 451.0] | 337.2 [204.3 to 556.6] | 20.0 [20.0 to 20.0]
  ST5 Day 365 | 52.9 [37.7 to 74.4] | 43.8 [29.7 to 64.6] | 20.0 [20.0 to 20.0]
  ST5 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST5 Day 545 | 31.0 [23.9 to 40.3] | 27.6 [21.7 to 35.0] | 20.0 [20.0 to 20.0]
  ST6 Day 1 | 21.8 [19.3 to 24.8] | 20.9 [19.1 to 22.8] | 21.7 [18.1 to 26.1]
  ST6 Day 29 | 22.0 [19.2 to 25.1] | 21.5 [19.4 to 23.8] | 21.3 [18.6 to 24.3]
  ST6 Day 57 | 22.7 [19.6 to 26.4] | 21.7 [19.3 to 24.3] | 21.7 [18.2 to 25.9]
  ST6 Day 85 | 69.0 [46.8 to 101.9] | 82.1 [56.8 to 118.7] | 20.0 [20.0 to 20.0]
  ST6 Day 180 | 32.3 [25.2 to 41.4] | 31.6 [25.0 to 39.9] | 21.9 [18.0 to 26.7]
  ST6 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST6 Day 208 | 305.1 [188.3 to 494.3] | 361.4 [225.9 to 578.3] | 21.8 [18.0 to 26.4]
  ST6 Day 365 | 60.7 [42.0 to 87.9] | 56.6 [38.3 to 83.7] | 21.4 [18.5 to 24.6]
  ST6 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST6 Day 545 | 30.9 [23.5 to 40.8] | 31.6 [24.1 to 41.4] | 20.0 [20.0 to 20.0]

7. Secondary Outcome: SCR for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 18 - 49 Years
Description: SCR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 18 - 49 years. Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): >=4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 55 | 57 | 30
Percentage of Participants
  ST1 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST1 Day 29 | 1.9 [0.3 to 9.9] | 1.8 [0.3 to 9.3] | 0.0 [0.0 to 11.4]
  ST1 Day 57 | 5.5 [1.9 to 14.9] | 3.5 [1.0 to 11.9] | 0.0 [0.0 to 11.4]
  ST1 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST1 Day 85 | 54.7 [41.5 to 67.3] | 70.9 [57.9 to 81.2] | 3.3 [0.6 to 16.7]
  ST1 Day 180 | 18.2 [10.2 to 30.3] | 19.3 [11.1 to 31.3] | 6.7 [1.8 to 21.3]
  ST1 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST1 Day 208 | 93.9 [83.5 to 97.9] | 94.2 [84.4 to 98.0] | 0.0 [0.0 to 12.9]
  ST1 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST1 Day 365 | 51.9 [38.7 to 64.9] | 38.0 [25.9 to 51.8] | 3.4 [0.6 to 17.2]
  ST1 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST1 Day 545 | 20.0 [10.9 to 33.8] | 12.2 [5.3 to 25.5] | 0.0 [0.0 to 12.9]
  ST2 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST2 Day 29 | 3.8 [1.0 to 12.8] | 5.3 [1.8 to 14.4] | 0.0 [0.0 to 11.4]
  ST2 Day 57 | 1.8 [0.3 to 9.6] | 7.0 [2.8 to 16.7] | 0.0 [0.0 to 11.4]
  ST2 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST2 Day 85 | 84.9 [72.9 to 92.1] | 90.9 [80.4 to 96.1] | 0.0 [0.0 to 11.4]
  ST2 Day 180 | 34.5 [23.4 to 47.7] | 38.6 [27.1 to 51.6] | 0.0 [0.0 to 11.4]
  ST2 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST2 Day 208 | 100 [92.7 to 100] | 100 [93.1 to 100] | 0.0 [0.0 to 12.9]
  ST2 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST2 Day 365 | 73.1 [59.7 to 83.2] | 70.0 [56.2 to 80.9] | 0.0 [0.0 to 11.7]
  ST2 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST2 Day 545 | 53.3 [39.1 to 67.1] | 36.6 [23.6 to 51.9] | 3.8 [0.7 to 18.9]
  ST3 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST3 Day 29 | 3.8 [1.0 to 12.8] | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 11.4]
  ST3 Day 57 | 1.8 [0.3 to 9.6] | 1.8 [0.3 to 9.3] | 0.0 [0.0 to 11.4]
  ST3 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST3 Day 85 | 84.9 [72.9 to 92.1] | 92.7 [82.7 to 97.1] | 3.3 [0.6 to 16.7]
  ST3 Day 180 | 41.8 [29.7 to 55.0] | 52.6 [39.9 to 65.0] | 3.3 [0.6 to 16.7]
  ST3 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST3 Day 208 | 100 [92.7 to 100] | 100 [93.1 to 100] | 0.0 [0.0 to 12.9]
  ST3 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST3 Day 365 | 69.2 [55.7 to 80.1] | 72.0 [58.3 to 82.5] | 0.0 [0.0 to 11.7]
  ST3 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST3 Day 545 | 42.2 [29.0 to 56.7] | 39.0 [25.7 to 54.3] | 0.0 [0.0 to 12.9]
  ST4 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST4 Day 29 | 1.9 [0.3 to 9.9] | 1.8 [0.3 to 9.3] | 0.0 [0.0 to 11.4]
  ST4 Day 57 | 1.8 [0.3 to 9.6] | 3.5 [1.0 to 11.9] | 6.7 [1.8 to 21.3]
  ST4 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST4 Day 85 | 75.5 [62.4 to 85.1] | 87.3 [76.0 to 93.7] | 6.7 [1.8 to 21.3]
  ST4 Day 180 | 25.5 [15.8 to 38.3] | 24.6 [15.2 to 37.1] | 6.7 [1.8 to 21.3]
  ST4 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST4 Day 208 | 100 [92.7 to 100] | 100 [93.1 to 100] | 7.7 [2.1 to 24.1]
  ST4 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST4 Day 365 | 61.5 [48.0 to 73.5] | 52.0 [38.5 to 65.2] | 3.4 [0.6 to 17.2]
  ST4 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST4 Day 545 | 46.7 [32.9 to 60.9] | 29.3 [17.6 to 44.5] | 7.7 [2.1 to 24.1]
  ST5 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST5 Day 29 | 1.9 [0.3 to 9.9] | 1.8 [0.3 to 9.3] | 0.0 [0.0 to 11.4]
  ST5 Day 57 | 1.8 [0.3 to 9.6] | 3.5 [1.0 to 11.9] | 0.0 [0.0 to 11.4]
  ST5 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST5 Day 85 | 73.6 [60.4 to 83.6] | 81.8 [69.7 to 89.8] | 0.0 [0.0 to 11.4]
  ST5 Day 180 | 21.8 [12.9 to 34.4] | 26.3 [16.6 to 39.0] | 0.0 [0.0 to 11.4]
  ST5 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST5 Day 208 | 95.9 [86.3 to 98.9] | 98.1 [89.9 to 99.7] | 0.0 [0.0 to 12.9]
  ST5 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST5 Day 365 | 51.9 [38.7 to 64.9] | 48.0 [34.8 to 61.5] | 0.0 [0.0 to 11.7]
  ST5 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST5 Day 545 | 37.8 [25.1 to 52.4] | 26.8 [15.7 to 41.9] | 3.8 [0.7 to 18.9]
  ST6 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST6 Day 29 | 3.8 [1.0 to 12.8] | 1.8 [0.3 to 9.3] | 0.0 [0.0 to 11.4]
  ST6 Day 57 | 3.6 [1.0 to 12.3] | 7.0 [2.8 to 16.7] | 3.3 [0.6 to 16.7]
  ST6 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST6 Day 85 | 62.3 [48.8 to 74.1] | 70.9 [57.9 to 81.2] | 0.0 [0.0 to 11.4]
  ST6 Day 180 | 25.5 [15.8 to 38.3] | 22.8 [13.8 to 35.2] | 3.3 [0.6 to 16.7]
  ST6 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST6 Day 208 | 89.8 [78.2 to 95.6] | 96.2 [87.0 to 98.9] | 0.0 [0.0 to 12.9]
  ST6 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST6 Day 365 | 55.8 [42.3 to 68.4] | 44.0 [31.2 to 57.7] | 3.4 [0.6 to 17.2]
  ST6 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST6 Day 545 | 37.8 [25.1 to 52.4] | 14.6 [6.9 to 28.4] | 0.0 [0.0 to 12.9]

8. Secondary Outcome: SCR for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 50 - 65 Years
Description: SCR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 50 - 65 years. Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): >=4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 30 | 29 | 13
Percentage of Participants
  ST1 Day 29 | 3.3 [0.6 to 16.7] | 0.0 [0.0 to 11.7] | 7.7 [1.4 to 33.3]
  ST1 Day 57 | 3.3 [0.6 to 16.7] | 3.4 [0.6 to 17.2] | 0.0 [0.0 to 22.8]
  ST1 Day 85 | 66.7 [48.8 to 80.8] | 65.5 [47.3 to 80.1] | 0.0 [0.0 to 22.8]
  ST1 Day 180 | 6.7 [1.8 to 21.3] | 20.7 [9.8 to 38.4] | 0.0 [0.0 to 22.8]
  ST1 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST1 Day 208 | 89.7 [73.6 to 96.4] | 92.9 [77.4 to 98.0] | 0.0 [0.0 to 24.2]
  ST1 Day 365 | 46.7 [30.2 to 63.9] | 37.9 [22.7 to 56.0] | 0.0 [0.0 to 22.8]
  ST1 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST1 Day 545 | 14.3 [5.7 to 31.5] | 16.7 [6.7 to 35.9] | 0.0 [0.0 to 24.2]
  ST2 Day 29 | 0.0 [0.0 to 11.4] | 6.9 [1.9 to 22.0] | 0.0 [0.0 to 22.8]
  ST2 Day 57 | 0.0 [0.0 to 11.4] | 3.4 [0.6 to 17.2] | 0.0 [0.0 to 22.8]
  ST2 Day 85 | 83.3 [66.4 to 92.7] | 86.2 [69.4 to 94.5] | 0.0 [0.0 to 22.8]
  ST2 Day 180 | 30.0 [16.7 to 47.9] | 37.9 [22.7 to 56.0] | 0.0 [0.0 to 22.8]
  ST2 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST2 Day 208 | 89.7 [73.6 to 96.4] | 96.4 [82.3 to 99.4] | 0.0 [0.0 to 24.2]
  ST2 Day 365 | 70.0 [52.1 to 83.3] | 72.4 [54.3 to 85.3] | 0.0 [0.0 to 22.8]
  ST2 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST2 Day 545 | 32.1 [17.9 to 50.7] | 33.3 [18.0 to 53.3] | 0.0 [0.0 to 24.2]
  ST3 Day 29 | 3.3 [0.6 to 16.7] | 0.0 [0.0 to 11.7] | 0.0 [0.0 to 22.8]
  ST3 Day 57 | 3.3 [0.6 to 16.7] | 0.0 [0.0 to 11.7] | 0.0 [0.0 to 22.8]
  ST3 Day 85 | 83.3 [66.4 to 92.7] | 89.7 [73.6 to 96.4] | 0.0 [0.0 to 22.8]
  ST3 Day 180 | 36.7 [21.9 to 54.5] | 44.8 [28.4 to 62.5] | 0.0 [0.0 to 22.8]
  ST3 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST3 Day 208 | 96.6 [82.8 to 99.4] | 92.9 [77.4 to 98.0] | 0.0 [0.0 to 24.2]
  ST3 Day 365 | 73.3 [55.6 to 85.8] | 69.0 [50.8 to 82.7] | 0.0 [0.0 to 22.8]
  ST3 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST3 Day 545 | 42.9 [26.5 to 60.9] | 33.3 [18.0 to 53.3] | 0.0 [0.0 to 24.2]
  ST4 Day 29 | 0.0 [0.0 to 11.4] | 0.0 [0.0 to 11.7] | 7.7 [1.4 to 33.3]
  ST4 Day 57 | 3.3 [0.6 to 16.7] | 0.0 [0.0 to 11.7] | 0.0 [0.0 to 22.8]
  ST4 Day 85 | 73.3 [55.6 to 85.8] | 75.9 [57.9 to 87.8] | 7.7 [1.4 to 33.3]
  ST4 Day 180 | 26.7 [14.2 to 44.4] | 24.1 [12.2 to 42.1] | 0.0 [0.0 to 22.8]
  ST4 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST4 Day 208 | 93.1 [78.0 to 98.1] | 96.4 [82.3 to 99.4] | 0.0 [0.0 to 24.2]
  ST4 Day 365 | 63.3 [45.5 to 78.1] | 51.7 [34.4 to 68.6] | 0.0 [0.0 to 22.8]
  ST4 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST4 Day 545 | 28.6 [15.3 to 47.1] | 25.0 [12.0 to 44.9] | 0.0 [0.0 to 24.2]
  ST5 Day 29 | 0.0 [0.0 to 11.4] | 6.9 [1.9 to 22.0] | 0.0 [0.0 to 22.8]
  ST5 Day 57 | 0.0 [0.0 to 11.4] | 6.9 [1.9 to 22.0] | 0.0 [0.0 to 22.8]
  ST5 Day 85 | 73.3 [55.6 to 85.8] | 79.3 [61.6 to 90.2] | 0.0 [0.0 to 22.8]
  ST5 Day 180 | 16.7 [7.3 to 33.6] | 24.1 [12.2 to 42.1] | 0.0 [0.0 to 22.8]
  ST5 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST5 Day 208 | 93.1 [78.0 to 98.1] | 92.9 [77.4 to 98.0] | 0.0 [0.0 to 24.2]
  ST5 Day 365 | 56.7 [39.2 to 72.6] | 48.3 [31.4 to 65.6] | 0.0 [0.0 to 22.8]
  ST5 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST5 Day 545 | 28.6 [15.3 to 47.1] | 29.2 [14.9 to 49.2] | 0.0 [0.0 to 24.2]
  ST6 Day 29 | 0.0 [0.0 to 11.4] | 3.4 [0.6 to 17.2] | 7.7 [1.4 to 33.3]
  ST6 Day 57 | 3.3 [0.6 to 16.7] | 3.4 [0.6 to 17.2] | 7.7 [1.4 to 33.3]
  ST6 Day 85 | 60.0 [42.3 to 75.4] | 72.4 [54.3 to 85.3] | 0.0 [0.0 to 22.8]
  ST6 Day 180 | 30.0 [16.7 to 47.9] | 34.5 [19.9 to 52.7] | 7.7 [1.4 to 33.3]
  ST6 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST6 Day 208 | 89.7 [73.6 to 96.4] | 96.4 [82.3 to 99.4] | 8.3 [1.5 to 35.4]
  ST6 Day 365 | 56.7 [39.2 to 72.6] | 58.6 [40.7 to 74.5] | 7.7 [1.4 to 33.3]
  ST6 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST6 Day 545 | 21.4 [10.2 to 39.5] | 33.3 [18.0 to 53.3] | 0.0 [0.0 to 24.2]

9. Secondary Outcome: GMFRs for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 18 - 49 Years
Description: GMFR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 18 - 49 years.
Time Frame: Day 1 (baseline), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12) and Day 545 (Month 18)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 55 | 57 | 30
Fold Rise
  ST1 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST1 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST1 Day 57 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST1 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST1 Day 85 | 2.9 [2.1 to 4.1] | 4.1 [3.0 to 5.6] | 1.0 [0.9 to 1.1]
  ST1 Day 180 | 1.3 [1.1 to 1.6] | 1.2 [1.1 to 1.4] | 1.0 [0.9 to 1.1]
  ST1 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST1 Day 208 | 13.6 [9.7 to 19.2] | 14.3 [10.4 to 19.7] | 1.0 [0.9 to 1.0]
  ST1 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST1 Day 365 | 2.3 [1.8 to 3.0] | 1.8 [1.5 to 2.3] | 1.0 [0.9 to 1.1]
  ST1 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST1 Day 545 | 1.5 [1.1 to 1.9] | 1.1 [1.0 to 1.3] | 0.9 [0.8 to 1.0]
  ST2 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST2 Day 29 | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.3] | 1.0 [1.0 to 1.0]
  ST2 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST2 Day 85 | 7.6 [5.5 to 10.5] | 9.8 [7.2 to 13.1] | 1.0 [1.0 to 1.0]
  ST2 Day 180 | 1.8 [1.4 to 2.3] | 1.8 [1.5 to 2.2] | 1.0 [1.0 to 1.0]
  ST2 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST2 Day 208 | 27.0 [20.5 to 35.5] | 29.1 [23.3 to 36.3] | 1.0 [1.0 to 1.0]
  ST2 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST2 Day 365 | 4.0 [3.0 to 5.4] | 3.3 [2.6 to 4.3] | 1.0 [1.0 to 1.0]
  ST2 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST2 Day 545 | 2.3 [1.7 to 2.9] | 1.6 [1.3 to 2.0] | 1.1 [0.9 to 1.3]
  ST3 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST3 Day 29 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST3 Day 57 | 1.0 [1.0 to 1.1] | 1.1 [0.9 to 1.2] | 1.0 [1.0 to 1.0]
  ST3 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST3 Day 85 | 8.7 [6.2 to 12.2] | 11.7 [8.6 to 15.8] | 1.1 [0.9 to 1.2]
  ST3 Day 180 | 2.0 [1.5 to 2.5] | 2.1 [1.7 to 2.6] | 1.0 [1.0 to 1.1]
  ST3 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST3 Day 208 | 28.1 [21.1 to 37.3] | 31.7 [25.4 to 39.5] | 1.0 [1.0 to 1.0]
  ST3 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST3 Day 365 | 3.9 [2.9 to 5.2] | 3.6 [2.7 to 4.6] | 1.0 [1.0 to 1.0]
  ST3 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST3 Day 545 | 2.0 [1.5 to 2.7] | 1.7 [1.4 to 2.1] | 1.0 [1.0 to 1.0]
  ST4 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST4 Day 29 | 1.0 [0.9 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST4 Day 57 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1]
  ST4 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST4 Day 85 | 4.0 [3.0 to 5.4] | 5.5 [4.2 to 7.1] | 1.0 [1.0 to 1.1]
  ST4 Day 180 | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.6] | 1.1 [1.0 to 1.1]
  ST4 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST4 Day 208 | 17.2 [13.0 to 22.9] | 19.1 [15.3 to 24.0] | 1.1 [1.0 to 1.1]
  ST4 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST4 Day 365 | 2.6 [2.0 to 3.4] | 2.1 [1.7 to 2.6] | 1.0 [1.0 to 1.1]
  ST4 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST4 Day 545 | 1.9 [1.5 to 2.5] | 1.4 [1.2 to 1.6] | 1.1 [0.9 to 1.4]
  ST5 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST5 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST5 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST5 Day 85 | 4.3 [3.2 to 5.8] | 5.3 [4.1 to 7.0] | 1.0 [1.0 to 1.0]
  ST5 Day 180 | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.6] | 1.0 [1.0 to 1.0]
  ST5 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST5 Day 208 | 16.9 [12.6 to 22.8] | 18.5 [14.4 to 23.9] | 1.0 [1.0 to 1.0]
  ST5 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST5 Day 365 | 2.6 [1.9 to 3.4] | 2.1 [1.7 to 2.7] | 1.0 [1.0 to 1.0]
  ST5 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST5 Day 545 | 1.8 [1.4 to 2.3] | 1.3 [1.1 to 1.6] | 1.0 [1.0 to 1.1]
  ST6 Day 29: number analyzed (Participants) | 53 | 57 | 30
  ST6 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST6 Day 57 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.1]
  ST6 Day 85: number analyzed (Participants) | 53 | 55 | 30
  ST6 Day 85 | 3.7 [2.7 to 5.1] | 4.2 [3.1 to 5.5] | 1.0 [1.0 to 1.0]
  ST6 Day 180 | 1.4 [1.2 to 1.8] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.1]
  ST6 Day 208: number analyzed (Participants) | 49 | 52 | 26
  ST6 Day 208 | 15.5 [11.1 to 21.4] | 16.4 [12.5 to 21.4] | 1.0 [1.0 to 1.0]
  ST6 Day 365: number analyzed (Participants) | 52 | 50 | 29
  ST6 Day 365 | 2.6 [1.9 to 3.6] | 2.0 [1.6 to 2.5] | 1.0 [1.0 to 1.1]
  ST6 Day 545: number analyzed (Participants) | 45 | 41 | 26
  ST6 Day 545 | 1.7 [1.3 to 2.3] | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]

10. Secondary Outcome: GMFRs for IgG Against Each OspA Serotype Stratified by Age Group During Main Study Phase: Group 50 - 65 Years
Description: GMFR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12) and 545 (Month 18) stratified by age group: 50 - 65 years.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 30 | 29 | 13
Fold Rise
  ST1 Day 29 | 1.0 [0.9 to 1.1] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2]
  ST1 Day 57 | 1.0 [0.9 to 1.1] | 1.1 [0.9 to 1.2] | 1.0 [1.0 to 1.0]
  ST1 Day 85 | 3.2 [2.3 to 4.5] | 3.1 [2.1 to 4.4] | 1.0 [0.9 to 1.0]
  ST1 Day 180 | 1.1 [1.0 to 1.3] | 1.2 [1.0 to 1.4] | 1.0 [0.9 to 1.0]
  ST1 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST1 Day 208 | 11.9 [7.2 to 19.5] | 12.3 [7.3 to 20.9] | 0.9 [0.8 to 1.1]
  ST1 Day 365 | 2.2 [1.5 to 3.1] | 1.8 [1.3 to 2.7] | 0.9 [0.8 to 1.1]
  ST1 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST1 Day 545 | 1.2 [1.0 to 1.5] | 1.2 [1.0 to 1.5] | 0.9 [0.8 to 1.1]
  ST2 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.3] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2] | 1.0 [1.0 to 1.0]
  ST2 Day 85 | 8.1 [5.3 to 12.5] | 8.2 [5.4 to 12.3] | 1.0 [1.0 to 1.0]
  ST2 Day 180 | 1.9 [1.3 to 2.8] | 1.7 [1.3 to 2.3] | 1.0 [1.0 to 1.0]
  ST2 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST2 Day 208 | 24.6 [15.1 to 40.0] | 28.8 [17.0 to 48.9] | 1.0 [1.0 to 1.0]
  ST2 Day 365 | 4.4 [2.9 to 6.9] | 4.0 [2.6 to 6.2] | 1.0 [1.0 to 1.0]
  ST2 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST2 Day 545 | 1.9 [1.3 to 2.8] | 1.7 [1.2 to 2.5] | 1.0 [1.0 to 1.0]
  ST3 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST3 Day 57 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST3 Day 85 | 7.4 [4.8 to 11.2] | 9.5 [6.4 to 14.3] | 1.0 [1.0 to 1.0]
  ST3 Day 180 | 1.7 [1.3 to 2.3] | 1.9 [1.4 to 2.6] | 1.0 [1.0 to 1.0]
  ST3 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST3 Day 208 | 22.0 [14.1 to 34.5] | 26.7 [15.4 to 46.5] | 1.0 [1.0 to 1.0]
  ST3 Day 365 | 3.8 [2.6 to 5.6] | 4.0 [2.6 to 6.2] | 1.0 [1.0 to 1.0]
  ST3 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST3 Day 545 | 1.8 [1.4 to 2.5] | 1.5 [1.2 to 2.0] | 1.0 [1.0 to 1.0]
  ST4 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2]
  ST4 Day 57 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST4 Day 85 | 3.6 [2.5 to 5.0] | 4.1 [2.9 to 5.9] | 1.1 [0.9 to 1.2]
  ST4 Day 180 | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.5] | 1.0 [1.0 to 1.0]
  ST4 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST4 Day 208 | 14.2 [9.0 to 22.4] | 16.2 [9.9 to 26.7] | 1.0 [1.0 to 1.0]
  ST4 Day 365 | 2.6 [1.8 to 3.6] | 2.2 [1.5 to 3.2] | 1.0 [1.0 to 1.0]
  ST4 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST4 Day 545 | 1.4 [1.1 to 1.8] | 1.3 [1.1 to 1.6] | 1.0 [1.0 to 1.0]
  ST5 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.3] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST5 Day 85 | 3.9 [2.7 to 5.6] | 4.5 [3.1 to 6.4] | 1.0 [1.0 to 1.0]
  ST5 Day 180 | 1.3 [1.0 to 1.6] | 1.3 [1.1 to 1.6] | 1.0 [1.0 to 1.0]
  ST5 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST5 Day 208 | 14.0 [9.3 to 21.2] | 16.9 [10.2 to 27.8] | 1.0 [1.0 to 1.0]
  ST5 Day 365 | 2.5 [1.8 to 3.5] | 2.2 [1.5 to 3.2] | 1.0 [1.0 to 1.0]
  ST5 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST5 Day 545 | 1.5 [1.2 to 1.9] | 1.4 [1.1 to 1.8] | 1.0 [1.0 to 1.0]
  ST6 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [0.8 to 1.2]
  ST6 Day 57 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [0.8 to 1.3]
  ST6 Day 85 | 3.2 [2.2 to 4.5] | 3.9 [2.7 to 5.7] | 0.9 [0.8 to 1.1]
  ST6 Day 180 | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 1.9] | 1.0 [0.8 to 1.3]
  ST6 Day 208: number analyzed (Participants) | 29 | 28 | 12
  ST6 Day 208 | 13.9 [8.7 to 22.2] | 17.3 [10.7 to 28.0] | 1.0 [0.7 to 1.3]
  ST6 Day 365 | 2.8 [1.9 to 4.0] | 2.7 [1.8 to 4.0] | 1.0 [0.8 to 1.2]
  ST6 Day 545: number analyzed (Participants) | 28 | 24 | 12
  ST6 Day 545 | 1.4 [1.1 to 1.8] | 1.5 [1.2 to 2.0] | 0.9 [0.7 to 1.1]

11. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) During the Main Study Phase
Description: SAE was any untoward medical occurrence that at any dose resulted in any of the following outcomes or deemed significant for any other reason: death; required inpatient prolonged existing hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 4.1 [1.6 to 10.1] | 4.1 [1.6 to 10.0] | 3.9 [1.1 to 13.2]

12. Secondary Outcome: Percentage of Participants With Related SAEs During the Main Study Phase
Description: SAE was any untoward medical occurrence that at any dose resulted in any of the following outcomes or deemed significant for any other reason: death; required inpatient prolonged existing hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to study vaccine was assessed by the investigator. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 7.0]

13. Secondary Outcome: Percentage of Participants Adverse Event of Special Interest (AESIs) During the Main Study Phase
Description: AESIs were defined as serious or non-serious AEs which were of scientific and medical concern specific to the investigational product. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 2.1 [0.6 to 7.2] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 7.0]

14. Secondary Outcome: Percentage of Participants With Related AESIs During the Main Study Phase
Description: AESIs were defined as serious or non-serious AEs which were of scientific and medical concern specific to the investigational product. Relatedness to study vaccine was assessed by the investigator. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 1.0 [0.2 to 5.6] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 7.0]

15. Secondary Outcome: Percentage of Participants With Unsolicited AEs During the Main Study Phase
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant temporally associated with the use of investigational product, whether or not related to investigational product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up (more than 6 days after vaccination) for solicited symptoms. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 66.0 [56.1 to 74.6] | 64.3 [54.4 to 73.1] | 68.6 [55.0 to 79.7]

16. Secondary Outcome: Percentage of Participants With Related Unsolicited AEs During the Main Study Phase
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant temporally associated with the use of investigational product, whether or not related to investigational product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up (more than 6 days after vaccination) for solicited symptoms. Relatedness to study vaccine was assessed by the investigator. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants | 18.6 [12.1 to 27.4] | 22.4 [15.3 to 31.7] | 7.8 [3.1 to 18.5]

17. Secondary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Each and After Any Vaccination During the Main Study Phase
Description: Solicited local AEs included pain, tenderness, induration (hardening), swelling and erythema (redness). Solicited systemic AEs included headache, myalgia (muscle pain), arthralgia (joint pain), fever (oral body temperature), flu-like symptoms, nausea, vomiting and fatigue. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: Up to 7 days after Vaccination 1, 2 and 3; Up to 7 days after any vaccination
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants
  Any solicited local AE: Any vaccination | 95.9 [89.9 to 98.4] | 98.0 [92.9 to 99.4] | 45.1 [32.3 to 58.6]
  Solicited local AE: 1st vaccination | 94.8 [88.5 to 97.8] | 93.9 [87.3 to 97.2] | 25.5 [15.5 to 38.9]
  Solicited local AE: 2nd vaccination | 80.4 [71.4 to 87.1] | 83.7 [75.1 to 89.7] | 23.5 [14.0 to 36.8]
  Solicited local AE: 3rd vaccination | 78.4 [69.2 to 85.4] | 82.7 [74.0 to 88.9] | 17.6 [9.6 to 30.3]
  Any solicited systemic AE: Any vaccination | 78.4 [69.2 to 85.4] | 69.4 [59.7 to 77.6] | 51.0 [37.7 to 64.1]
  Solicited systemic AE: 1st vaccination | 61.9 [51.9 to 70.9] | 56.1 [46.3 to 65.5] | 35.3 [23.6 to 49.0]
  Solicited systemic AE: 2nd vaccination | 47.4 [37.8 to 57.3] | 40.8 [31.6 to 50.7] | 21.6 [12.5 to 34.6]
  Solicited systemic AE: 3rd vaccination | 36.1 [27.2 to 46.0] | 40.8 [31.6 to 50.7] | 17.6 [9.6 to 30.3]

18. Secondary Outcome: Percentage of Participants With SAEs, AESIs, Solicited and Unsolicited AEs Stratified by Age Group During the Main Study Phase
Description: Percentage of participants with SAEs, AESIs, solicited and unsolicited AEs during main study phase stratified by age group 18-49 years and 50-65 years were reported. SAE: any untoward medical occurrence that at any dose resulted in any of the following outcomes or deemed significant for any other reason: death; required inpatient prolonged existing hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect. AESI: any AEs of scientific/medical concern specific to study vaccine. Solicited AE: predefined reactions at injection site or systemic reactions after each vaccination. Unsolicited AE: any untoward medical occurrence in participant associated with use of study vaccine, whether or not related to study vaccine, reported in addition to solicited and any solicited symptom with onset outside specified period of follow-up. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 545 (Month 18)
Population: Safety population included all participants who entered into the study and received at least 1 dose of vaccination. Here "Number Analyzed" signifies participants evaluable for this outcome measure at specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VLA15 With Alum Lower Dose | VLA15 With Alum Higher Dose | Placebo
Number analyzed (Participants) | 97 | 98 | 51
Percentage of Participants
  SAE: 18-49 Years: number analyzed (Participants) | 64 | 64 | 32
  SAE: 18-49 Years | 3.1 [0.9 to 10.7] | 3.1 [0.9 to 10.7] | 0.0 [0.0 to 10.7]
  SAE: 50-65 Years: number analyzed (Participants) | 33 | 34 | 19
  SAE: 50-65 Years | 6.1 [1.7 to 19.6] | 5.9 [1.6 to 19.1] | 10.5 [2.9 to 31.4]
  AESI: 18-49 Years: number analyzed (Participants) | 64 | 64 | 32
  AESI: 18-49 Years | 3.1 [0.9 to 10.7] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 10.7]
  AESI: 50-65 Years: number analyzed (Participants) | 33 | 34 | 19
  AESI: 50-65 Years | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.2] | 0.0 [0.0 to 16.8]
  Solicited AE: 18-49 Years: number analyzed (Participants) | 64 | 64 | 32
  Solicited AE: 18-49 Years | 95.3 [87.1 to 98.4] | 96.9 [89.3 to 99.1] | 59.4 [42.3 to 74.5]
  Solicited AE: 50-65 Years: number analyzed (Participants) | 33 | 34 | 19
  Solicited AE: 50-65 Years | 100 [89.6 to 100] | 100 [89.8 to 100] | 73.7 [51.2 to 88.2]
  Unsolicited AE: 18-49 Years: number analyzed (Participants) | 64 | 64 | 32
  Unsolicited AE: 18-49 Years | 64.1 [51.8 to 74.7] | 65.6 [53.4 to 76.1] | 59.4 [42.3 to 74.5]
  Unsolicited AE: 50-65 Years: number analyzed (Participants) | 33 | 34 | 19
  Unsolicited AE: 50-65 Years | 69.7 [52.7 to 82.6] | 61.8 [45.0 to 76.1] | 84.2 [62.4 to 94.5]

19. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6): Booster Per-protocol (PP) Population
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24, and Month 30. The outcome measure was planned to be analyzed for Booster PP population from Day 1 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: At Day 1 (Month 0), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12), Day 545 (Month 18), Month 19, Month 24, and Month 30
Population: Booster per-protocol (PP) population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity) and who were enrolled into the booster phase despite exclusion from the PP population of main study phase. Here, "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 37 | 18
Units per milliliter (U/mL)
  ST1 Day 1 | 20.5 [19.5 to 21.4] | 20.0 [20.0 to 20.0]
  ST1 Day 29 | 20.9 [19.6 to 22.3] | 20.0 [20.0 to 20.0]
  ST1 Day 57 | 22.6 [19.8 to 25.8] | 20.0 [20.0 to 20.0]
  ST1 Day 85: number analyzed (Participants) | 37 | 17
  ST1 Day 85 | 78.9 [53.2 to 117.1] | 67.2 [41.2 to 109.6]
  ST1 Day 180 | 27.6 [23.4 to 32.5] | 24.2 [19.4 to 30.3]
  ST1 Day 208: number analyzed (Participants) | 35 | 17
  ST1 Day 208 | 292.0 [198.1 to 430.3] | 349.5 [184.4 to 662.4]
  ST1 Day 365: number analyzed (Participants) | 37 | 17
  ST1 Day 365 | 39.7 [30.0 to 52.4] | 37.3 [20.9 to 66.4]
  ST1 Day 545 | 24.9 [21.2 to 29.2] | 24.0 [17.9 to 32.3]
  ST1 Month 19 | 1277.0 [861.8 to 1892.3] | 23.6 [18.1 to 30.8]
  ST1 Month 24: number analyzed (Participants) | 37 | 17
  ST1 Month 24 | 137.4 [95.8 to 196.9] | 22.3 [17.7 to 28.0]
  ST1 Month 30: number analyzed (Participants) | 37 | 17
  ST1 Month 30 | 54.1 [38.6 to 75.7] | 22.1 [17.9 to 27.4]
  ST2 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29 | 23.4 [20.0 to 27.2] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 23.2 [19.3 to 27.8] | 20.0 [20.0 to 20.0]
  ST2 Day 85: number analyzed (Participants) | 37 | 17
  ST2 Day 85 | 219.3 [156.5 to 307.4] | 187.4 [109.2 to 321.8]
  ST2 Day 180 | 41.0 [31.1 to 54.1] | 33.5 [22.9 to 48.8]
  ST2 Day 208: number analyzed (Participants) | 35 | 17
  ST2 Day 208 | 606.3 [419.0 to 877.3] | 694.7 [427.9 to 1127.9]
  ST2 Day 365: number analyzed (Participants) | 37 | 17
  ST2 Day 365 | 76.1 [55.0 to 105.5] | 75.5 [44.0 to 129.6]
  ST2 Day 545 | 31.8 [25.2 to 40.1] | 35.9 [25.2 to 51.2]
  ST2 Month 19 | 2194.5 [1566.8 to 3073.7] | 36.8 [26.4 to 51.3]
  ST2 Month 24: number analyzed (Participants) | 37 | 17
  ST2 Month 24 | 258.6 [197.4 to 338.8] | 26.0 [19.9 to 34.1]
  ST2 Month 30: number analyzed (Participants) | 37 | 17
  ST2 Month 30 | 89.5 [63.4 to 126.2] | 21.9 [18.0 to 26.6]
  ST3 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 21.8 [18.3 to 25.9] | 20.0 [20.0 to 20.0]
  ST3 Day 85: number analyzed (Participants) | 37 | 17
  ST3 Day 85 | 235.1 [155.9 to 354.3] | 237.6 [152.4 to 370.4]
  ST3 Day 180 | 47.6 [36.7 to 61.7] | 43.9 [28.0 to 68.8]
  ST3 Day 208: number analyzed (Participants) | 35 | 17
  ST3 Day 208 | 631.9 [431.2 to 925.9] | 666.3 [393.9 to 1127.3]
  ST3 Day 365: number analyzed (Participants) | 37 | 17
  ST3 Day 365 | 78.7 [57.2 to 108.3] | 81.1 [44.0 to 149.7]
  ST3 Day 545 | 31.1 [24.8 to 38.8] | 39.5 [25.9 to 60.4]
  ST3 Month 19 | 1916.2 [1320.7 to 2780.2] | 35.8 [24.9 to 51.7]
  ST3 Month 24: number analyzed (Participants) | 37 | 17
  ST3 Month 24 | 265.8 [202.9 to 348.2] | 29.1 [20.8 to 40.6]
  ST3 Month 30: number analyzed (Participants) | 37 | 17
  ST3 Month 30 | 101.6 [77.6 to 133.1] | 24.9 [19.0 to 32.6]
  ST4 Day 1 | 20.8 [19.2 to 22.4] | 20.0 [20.0 to 20.0]
  ST4 Day 29 | 21.2 [19.5 to 23.1] | 20.0 [20.0 to 20.0]
  ST4 Day 57 | 22.2 [19.6 to 25.1] | 20.0 [20.0 to 20.0]
  ST4 Day 85: number analyzed (Participants) | 37 | 17
  ST4 Day 85 | 108.9 [75.9 to 156.3] | 100.7 [65.1 to 155.6]
  ST4 Day 180 | 30.1 [24.7 to 36.6] | 28.4 [21.2 to 38.2]
  ST4 Day 208: number analyzed (Participants) | 35 | 17
  ST4 Day 208 | 376.6 [261.1 to 543.3] | 455.3 [268.2 to 773.1]
  ST4 Day 365: number analyzed (Participants) | 37 | 17
  ST4 Day 365 | 47.5 [35.8 to 62.9] | 46.5 [26.7 to 80.9]
  ST4 Day 545 | 28.8 [23.8 to 34.8] | 31.3 [22.5 to 43.7]
  ST4 Month 19 | 1661.1 [1156.4 to 2386.0] | 26.5 [19.9 to 35.4]
  ST4 Month 24: number analyzed (Participants) | 37 | 17
  ST4 Month 24 | 200.7 [150.9 to 266.8] | 24.6 [18.9 to 32.0]
  ST4 Month 30: number analyzed (Participants) | 37 | 17
  ST4 Month 30 | 72.3 [52.2 to 100.1] | 22.1 [17.9 to 27.3]
  ST5 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29 | 22.1 [19.5 to 25.0] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 23.3 [19.7 to 27.5] | 20.0 [20.0 to 20.0]
  ST5 Day 85: number analyzed (Participants) | 37 | 17
  ST5 Day 85 | 100.9 [70.6 to 144.1] | 127.4 [85.5 to 189.8]
  ST5 Day 180 | 26.5 [22.3 to 31.6] | 32.3 [23.4 to 44.7]
  ST5 Day 208: number analyzed (Participants) | 35 | 17
  ST5 Day 208 | 370.6 [257.3 to 533.8] | 528.4 [330.8 to 844.0]
  ST5 Day 365: number analyzed (Participants) | 37 | 17
  ST5 Day 365 | 43.9 [32.5 to 59.3] | 59.4 [35.9 to 98.4]
  ST5 Day 545 | 25.0 [21.1 to 29.7] | 31.1 [22.0 to 44.0]
  ST5 Month 19 | 1507.9 [1066.0 to 2133.0] | 25.5 [19.2 to 33.8]
  ST5 Month 24: number analyzed (Participants) | 37 | 17
  ST5 Month 24 | 170.2 [127.2 to 227.7] | 23.7 [18.5 to 30.3]
  ST5 Month 30: number analyzed (Participants) | 37 | 17
  ST5 Month 30 | 74.0 [54.9 to 99.7] | 23.6 [18.6 to 29.9]
  ST6 Day 1 | 20.9 [19.2 to 22.7] | 20.0 [20.0 to 20.0]
  ST6 Day 29 | 22.0 [19.6 to 24.7] | 20.0 [20.0 to 20.0]
  ST6 Day 57 | 24.8 [20.7 to 29.9] | 20.0 [20.0 to 20.0]
  ST6 Day 85: number analyzed (Participants) | 37 | 17
  ST6 Day 85 | 82.0 [57.3 to 117.3] | 116.5 [74.3 to 182.5]
  ST6 Day 180 | 29.2 [23.8 to 35.7] | 36.4 [25.4 to 52.2]
  ST6 Day 208: number analyzed (Participants) | 35 | 17
  ST6 Day 208 | 351.9 [246.7 to 502.0] | 509.0 [308.6 to 839.4]
  ST6 Day 365: number analyzed (Participants) | 37 | 17
  ST6 Day 365 | 46.8 [33.7 to 65.0] | 67.3 [41.6 to 108.7]
  ST6 Day 545 | 26.3 [21.6 to 32.0] | 29.1 [21.0 to 40.4]
  ST6 Month 19 | 1406.8 [996.2 to 1986.7] | 28.7 [21.1 to 39.2]
  ST6 Month 24: number analyzed (Participants) | 37 | 17
  ST6 Month 24 | 181.5 [138.9 to 237.1] | 25.8 [19.9 to 33.5]
  ST6 Month 30: number analyzed (Participants) | 37 | 17
  ST6 Month 30 | 76.0 [55.7 to 103.8] | 23.8 [18.4 to 30.6]

20. Secondary Outcome: SCRs for Each OspA Serotype Specific IgG (ST1 to ST6): Booster PP Population
Description: SCR for each OspA serotype specific IgG ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24, and Month 30. Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): greater than or equal to (>=) 4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants. Percentages are based on the number of participants with non-missing observations. The outcome measure was planned to be analyzed for Booster PP population from Day 29 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12), Day 545 (Month 18), Month 19, Month 24, and Month 30
Population: Booster PP population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity) and who were enrolled into the booster phase despite exclusion from the PP population of main study phase. Here, "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 37 | 18
Percentage of Participants
  ST1 Day 29 | 2.7 [0.5 to 13.8] | 0.0 [0.0 to 17.6]
  ST1 Day 57 | 8.1 [2.8 to 21.3] | 0.0 [0.0 to 17.6]
  ST1 Day 85: number analyzed (Participants) | 37 | 17
  ST1 Day 85 | 64.9 [48.8 to 78.2] | 70.6 [46.9 to 86.7]
  ST1 Day 180 | 29.7 [17.5 to 45.8] | 16.7 [5.8 to 39.2]
  ST1 Day 208: number analyzed (Participants) | 35 | 17
  ST1 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST1 Day 365: number analyzed (Participants) | 37 | 17
  ST1 Day 365 | 43.2 [28.7 to 59.1] | 29.4 [13.3 to 53.1]
  ST1 Day 545 | 16.2 [7.7 to 31.1] | 11.1 [3.1 to 32.8]
  ST1 Month 19 | 100 [90.6 to 100] | 11.1 [3.1 to 32.8]
  ST1 Month 24: number analyzed (Participants) | 37 | 17
  ST1 Month 24 | 89.2 [75.3 to 95.7] | 5.9 [1.0 to 27.0]
  ST1 Month 30: number analyzed (Participants) | 37 | 17
  ST1 Month 30 | 56.8 [40.9 to 71.3] | 5.9 [1.0 to 27.0]
  ST2 Day 29 | 10.8 [4.3 to 24.7] | 0.0 [0.0 to 17.6]
  ST2 Day 57 | 8.1 [2.8 to 21.3] | 0.0 [0.0 to 17.6]
  ST2 Day 85: number analyzed (Participants) | 37 | 17
  ST2 Day 85 | 97.3 [86.2 to 99.5] | 88.2 [65.7 to 96.7]
  ST2 Day 180 | 48.6 [33.4 to 64.1] | 33.3 [16.3 to 56.3]
  ST2 Day 208: number analyzed (Participants) | 35 | 17
  ST2 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST2 Day 365: number analyzed (Participants) | 37 | 17
  ST2 Day 365 | 75.7 [59.9 to 86.6] | 70.6 [46.9 to 86.7]
  ST2 Day 545 | 35.1 [21.8 to 51.2] | 44.4 [24.6 to 66.3]
  ST2 Month 19 | 100 [90.6 to 100] | 50.0 [29.0 to 71.0]
  ST2 Month 24: number analyzed (Participants) | 37 | 17
  ST2 Month 24 | 100 [90.6 to 100] | 23.5 [9.6 to 47.3]
  ST2 Month 30: number analyzed (Participants) | 37 | 17
  ST2 Month 30 | 73.0 [57.0 to 84.6] | 5.9 [1.0 to 27.0]
  ST3 Day 29 | 0.0 [0.0 to 9.4] | 0.0 [0.0 to 17.6]
  ST3 Day 57 | 2.7 [0.5 to 13.8] | 0.0 [0.0 to 17.6]
  ST3 Day 85: number analyzed (Participants) | 37 | 17
  ST3 Day 85 | 89.2 [75.3 to 95.7] | 100 [81.6 to 100]
  ST3 Day 180 | 59.5 [43.5 to 73.7] | 50.0 [29.0 to 71.0]
  ST3 Day 208: number analyzed (Participants) | 35 | 17
  ST3 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST3 Day 365: number analyzed (Participants) | 37 | 17
  ST3 Day 365 | 73.0 [57.0 to 84.6] | 70.6 [46.9 to 86.7]
  ST3 Day 545 | 32.4 [19.6 to 48.5] | 44.4 [24.6 to 66.3]
  ST3 Month 19 | 100 [90.6 to 100] | 44.4 [24.6 to 66.3]
  ST3 Month 24: number analyzed (Participants) | 37 | 17
  ST3 Month 24 | 100 [90.6 to 100] | 29.4 [13.3 to 53.1]
  ST3 Month 30: number analyzed (Participants) | 37 | 17
  ST3 Month 30 | 89.2 [75.3 to 95.7] | 17.6 [6.2 to 41.0]
  ST4 Day 29 | 2.7 [0.5 to 13.8] | 0.0 [0.0 to 17.6]
  ST4 Day 57 | 5.4 [1.5 to 17.7] | 0.0 [0.0 to 17.6]
  ST4 Day 85: number analyzed (Participants) | 37 | 17
  ST4 Day 85 | 81.1 [65.8 to 90.5] | 88.2 [65.7 to 96.7]
  ST4 Day 180 | 32.4 [19.6 to 48.5] | 27.8 [12.5 to 50.9]
  ST4 Day 208: number analyzed (Participants) | 35 | 17
  ST4 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST4 Day 365: number analyzed (Participants) | 37 | 17
  ST4 Day 365 | 56.8 [40.9 to 71.3] | 52.9 [31.0 to 73.8]
  ST4 Day 545 | 29.7 [17.5 to 45.8] | 38.9 [20.3 to 61.4]
  ST4 Month 19 | 100 [90.6 to 100] | 22.2 [9.0 to 45.2]
  ST4 Month 24: number analyzed (Participants) | 37 | 17
  ST4 Month 24 | 100 [90.6 to 100] | 17.6 [6.2 to 41.0]
  ST4 Month 30: number analyzed (Participants) | 37 | 17
  ST4 Month 30 | 73.0 [57.0 to 84.6] | 5.9 [1.0 to 27.0]
  ST5 Day 29 | 8.1 [2.8 to 21.3] | 0.0 [0.0 to 17.6]
  ST5 Day 57 | 10.8 [4.3 to 24.7] | 0.0 [0.0 to 17.6]
  ST5 Day 85: number analyzed (Participants) | 37 | 17
  ST5 Day 85 | 78.4 [62.8 to 88.6] | 94.1 [73.0 to 99.0]
  ST5 Day 180 | 24.3 [13.4 to 40.1] | 38.9 [20.3 to 61.4]
  ST5 Day 208: number analyzed (Participants) | 35 | 17
  ST5 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST5 Day 365: number analyzed (Participants) | 37 | 17
  ST5 Day 365 | 48.6 [33.4 to 64.1] | 70.6 [46.9 to 86.7]
  ST5 Day 545 | 18.9 [9.5 to 34.2] | 33.3 [16.3 to 56.3]
  ST5 Month 19 | 100 [90.6 to 100] | 16.7 [5.8 to 39.2]
  ST5 Month 24: number analyzed (Participants) | 37 | 17
  ST5 Month 24 | 97.3 [86.2 to 99.5] | 11.8 [3.3 to 34.3]
  ST5 Month 30: number analyzed (Participants) | 37 | 17
  ST5 Month 30 | 81.1 [65.8 to 90.5] | 11.8 [3.3 to 34.3]
  ST6 Day 29 | 5.4 [1.5 to 17.7] | 0.0 [0.0 to 17.6]
  ST6 Day 57 | 13.5 [5.9 to 28.0] | 0.0 [0.0 to 17.6]
  ST6 Day 85: number analyzed (Participants) | 37 | 17
  ST6 Day 85 | 70.3 [54.2 to 82.5] | 88.2 [65.7 to 96.7]
  ST6 Day 180 | 27.0 [15.4 to 43.0] | 44.4 [24.6 to 66.3]
  ST6 Day 208: number analyzed (Participants) | 35 | 17
  ST6 Day 208 | 97.1 [85.5 to 99.5] | 100 [81.6 to 100]
  ST6 Day 365: number analyzed (Participants) | 37 | 17
  ST6 Day 365 | 45.9 [31.0 to 61.6] | 76.5 [52.7 to 90.4]
  ST6 Day 545 | 16.2 [7.7 to 31.1] | 27.8 [12.5 to 50.9]
  ST6 Month 19 | 100 [90.6 to 100] | 27.8 [12.5 to 50.9]
  ST6 Month 24: number analyzed (Participants) | 37 | 17
  ST6 Month 24 | 97.3 [86.2 to 99.5] | 23.5 [9.6 to 47.3]
  ST6 Month 30: number analyzed (Participants) | 37 | 17
  ST6 Month 30 | 73.0 [57.0 to 84.6] | 11.8 [3.3 to 34.3]

21. Secondary Outcome: GMFR as Compared to Baseline for IgG Against Each OspA Serotype (ST1 to ST6): Booster PP Population
Description: GMFR as compared to baseline for IgG against each Osp serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24 and Month 30 were reported in this outcome measure. The outcome measure was planned to be analyzed for Booster PP population from Day 1 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: Day 1 (baseline from where comparison was done), Day 29 (Month 1), Day 57 (Month 2), Day 85 (Month 3), Day 180 (Month 6), Day 208 (Month 7), Day 365 (Month 12), Day 545 (Month 18), Month 19, Month 24, and Month 30
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 37 | 18
Fold Rise
  ST1 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST1 Day 57 | 1.1 [1.0 to 1.3] | 1.0 [1.0 to 1.0]
  ST1 Day 85: number analyzed (Participants) | 37 | 17
  ST1 Day 85 | 3.9 [2.6 to 5.7] | 3.4 [2.1 to 5.5]
  ST1 Day 180 | 1.3 [1.2 to 1.6] | 1.2 [1.0 to 1.5]
  ST1 Day 208: number analyzed (Participants) | 35 | 17
  ST1 Day 208 | 14.2 [9.7 to 21.0] | 17.5 [9.2 to 33.1]
  ST1 Day 365: number analyzed (Participants) | 37 | 17
  ST1 Day 365 | 1.9 [1.5 to 2.6] | 1.9 [1.0 to 3.3]
  ST1 Day 545 | 1.2 [1.0 to 1.4] | 1.2 [0.9 to 1.6]
  ST1 Month 19 | 62.4 [42.6 to 91.4] | 1.2 [0.9 to 1.5]
  ST1 Month 24: number analyzed (Participants) | 37 | 17
  ST1 Month 24 | 6.7 [4.7 to 9.6] | 1.1 [0.9 to 1.4]
  ST1 Month 30: number analyzed (Participants) | 37 | 17
  ST1 Month 30 | 2.6 [1.9 to 3.7] | 1.1 [0.9 to 1.4]
  ST2 Day 29 | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]
  ST2 Day 85: number analyzed (Participants) | 37 | 17
  ST2 Day 85 | 11.0 [7.8 to 15.4] | 9.4 [5.5 to 16.1]
  ST2 Day 180 | 2.1 [1.6 to 2.7] | 1.7 [1.1 to 2.4]
  ST2 Day 208: number analyzed (Participants) | 35 | 17
  ST2 Day 208 | 30.3 [21.0 to 43.9] | 34.7 [21.4 to 56.4]
  ST2 Day 365: number analyzed (Participants) | 37 | 17
  ST2 Day 365 | 3.8 [2.7 to 5.3] | 3.8 [2.2 to 6.5]
  ST2 Day 545 | 1.6 [1.3 to 2.0] | 1.8 [1.3 to 2.6]
  ST2 Month 19 | 109.7 [78.3 to 153.7] | 1.8 [1.3 to 2.6]
  ST2 Month 24: number analyzed (Participants) | 37 | 17
  ST2 Month 24 | 12.9 [9.9 to 16.9] | 1.3 [1.0 to 1.7]
  ST2 Month 30: number analyzed (Participants) | 37 | 17
  ST2 Month 30 | 4.5 [3.2 to 6.3] | 1.1 [0.9 to 1.3]
  ST3 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  ST3 Day 57 | 1.1 [0.9 to 1.3] | 1.0 [1.0 to 1.0]
  ST3 Day 85: number analyzed (Participants) | 37 | 17
  ST3 Day 85 | 11.8 [7.8 to 17.7] | 11.9 [7.6 to 18.5]
  ST3 Day 180 | 2.4 [1.8 to 3.1] | 2.2 [1.4 to 3.4]
  ST3 Day 208: number analyzed (Participants) | 35 | 17
  ST3 Day 208 | 31.6 [21.6 to 46.3] | 33.3 [19.7 to 56.4]
  ST3 Day 365: number analyzed (Participants) | 37 | 17
  ST3 Day 365 | 3.9 [2.9 to 5.4] | 4.1 [2.2 to 7.5]
  ST3 Day 545 | 1.6 [1.2 to 1.9] | 2.0 [1.3 to 3.0]
  ST3 Month 19 | 95.8 [66.0 to 139.0] | 1.8 [1.2 to 2.6]
  ST3 Month 24: number analyzed (Participants) | 37 | 17
  ST3 Month 24 | 13.3 [10.1 to 17.4] | 1.5 [1.0 to 2.0]
  ST3 Month 30: number analyzed (Participants) | 37 | 17
  ST3 Month 30 | 5.1 [3.9 to 6.7] | 1.2 [0.9 to 1.6]
  ST4 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST4 Day 57 | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST4 Day 85: number analyzed (Participants) | 37 | 17
  ST4 Day 85 | 5.2 [3.7 to 7.4] | 5.0 [3.3 to 7.8]
  ST4 Day 180 | 1.4 [1.2 to 1.7] | 1.4 [1.1 to 1.9]
  ST4 Day 208: number analyzed (Participants) | 35 | 17
  ST4 Day 208 | 18.1 [12.6 to 25.9] | 22.8 [13.4 to 38.7]
  ST4 Day 365: number analyzed (Participants) | 37 | 17
  ST4 Day 365 | 2.3 [1.7 to 3.0] | 2.3 [1.3 to 4.0]
  ST4 Day 545 | 1.4 [1.2 to 1.6] | 1.6 [1.1 to 2.2]
  ST4 Month 19 | 79.9 [56.5 to 113.1] | 1.3 [1.0 to 1.8]
  ST4 Month 24: number analyzed (Participants) | 37 | 17
  ST4 Month 24 | 9.7 [7.3 to 12.8] | 1.2 [0.9 to 1.6]
  ST4 Month 30: number analyzed (Participants) | 37 | 17
  ST4 Month 30 | 3.5 [2.5 to 4.8] | 1.1 [0.9 to 1.4]
  ST5 Day 29 | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]
  ST5 Day 85: number analyzed (Participants) | 37 | 17
  ST5 Day 85 | 5.0 [3.5 to 7.2] | 6.4 [4.3 to 9.5]
  ST5 Day 180 | 1.3 [1.1 to 1.6] | 1.6 [1.2 to 2.2]
  ST5 Day 208: number analyzed (Participants) | 35 | 17
  ST5 Day 208 | 18.5 [12.9 to 26.7] | 26.4 [16.5 to 42.2]
  ST5 Day 365: number analyzed (Participants) | 37 | 17
  ST5 Day 365 | 2.2 [1.6 to 3.0] | 3.0 [1.8 to 4.9]
  ST5 Day 545 | 1.3 [1.1 to 1.5] | 1.6 [1.1 to 2.2]
  ST5 Month 19 | 75.4 [53.3 to 106.7] | 1.3 [1.0 to 1.7]
  ST5 Month 24: number analyzed (Participants) | 37 | 17
  ST5 Month 24 | 8.5 [6.4 to 11.4] | 1.2 [0.9 to 1.5]
  ST5 Month 30: number analyzed (Participants) | 37 | 17
  ST5 Month 30 | 3.7 [2.7 to 5.0] | 1.2 [0.9 to 1.5]
  ST6 Day 29 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST6 Day 57 | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0]
  ST6 Day 85: number analyzed (Participants) | 37 | 17
  ST6 Day 85 | 3.9 [2.8 to 5.6] | 5.8 [3.7 to 9.1]
  ST6 Day 180 | 1.4 [1.2 to 1.7] | 1.8 [1.3 to 2.6]
  ST6 Day 208: number analyzed (Participants) | 35 | 17
  ST6 Day 208 | 16.8 [11.8 to 24.0] | 25.4 [15.4 to 42.0]
  ST6 Day 365: number analyzed (Participants) | 37 | 17
  ST6 Day 365 | 2.2 [1.6 to 3.1] | 3.4 [2.1 to 5.4]
  ST6 Day 545 | 1.3 [1.1 to 1.5] | 1.5 [1.1 to 2.0]
  ST6 Month 19 | 67.5 [48.4 to 94.0] | 1.4 [1.1 to 2.0]
  ST6 Month 24: number analyzed (Participants) | 37 | 17
  ST6 Month 24 | 8.7 [6.7 to 11.4] | 1.3 [1.0 to 1.7]
  ST6 Month 30: number analyzed (Participants) | 37 | 17
  ST6 Month 30 | 3.6 [2.7 to 4.9] | 1.2 [0.9 to 1.5]

22. Secondary Outcome: GMFR as Compared to Day 208 for IgG Against Each OspA Serotype (ST1 to ST6): Booster PP Population
Description: GMFR as compared to Day 208 for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Month 19, Month 24 and Month 30. The outcome measure was planned to be analyzed for Booster PP population from Day 208 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: Day 208 (from where comparison was done), Month 19, Month 24 and Month 30
Population: Booster PP population, excluded those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity) and who were enrolled into the booster phase despite exclusion from the PP population of main study phase. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 35 | 17
Fold Rise
  ST1 Month 19 | 4.2 [3.4 to 5.2] | 0.1 [0.0 to 0.1]
  ST1 Month 24: number analyzed (Participants) | 35 | 16
  ST1 Month 24 | 0.5 [0.4 to 0.6] | 0.1 [0.0 to 0.1]
  ST1 Month 30: number analyzed (Participants) | 35 | 16
  ST1 Month 30 | 0.2 [0.1 to 0.2] | 0.1 [0.0 to 0.1]
  ST2 Month 19 | 3.5 [2.9 to 4.3] | 0.1 [0.0 to 0.1]
  ST2 Month 24: number analyzed (Participants) | 35 | 16
  ST2 Month 24 | 0.4 [0.3 to 0.5] | 0.0 [0.0 to 0.1]
  ST2 Month 30: number analyzed (Participants) | 35 | 16
  ST2 Month 30 | 0.1 [0.1 to 0.2] | 0.0 [0.0 to 0.0]
  ST3 Month 19 | 2.9 [2.3 to 3.5] | 0.1 [0.0 to 0.1]
  ST3 Month 24: number analyzed (Participants) | 35 | 16
  ST3 Month 24 | 0.4 [0.3 to 0.5] | 0.0 [0.0 to 0.1]
  ST3 Month 30: number analyzed (Participants) | 35 | 16
  ST3 Month 30 | 0.2 [0.1 to 0.2] | 0.0 [0.0 to 0.1]
  ST4 Month 19 | 4.2 [3.5 to 5.1] | 0.1 [0.0 to 0.1]
  ST4 Month 24: number analyzed (Participants) | 35 | 16
  ST4 Month 24 | 0.5 [0.4 to 0.7] | 0.1 [0.0 to 0.1]
  ST4 Month 30: number analyzed (Participants) | 35 | 16
  ST4 Month 30 | 0.2 [0.1 to 0.3] | 0.0 [0.0 to 0.1]
  ST5 Month 19 | 4.0 [3.3 to 4.8] | 0.0 [0.0 to 0.1]
  ST5 Month 24: number analyzed (Participants) | 35 | 16
  ST5 Month 24 | 0.5 [0.4 to 0.6] | 0.0 [0.0 to 0.1]
  ST5 Month 30: number analyzed (Participants) | 35 | 16
  ST5 Month 30 | 0.2 [0.1 to 0.3] | 0.0 [0.0 to 0.1]
  ST6 Month 19 | 3.9 [3.2 to 4.7] | 0.1 [0.0 to 0.1]
  ST6 Month 24: number analyzed (Participants) | 35 | 16
  ST6 Month 24 | 0.5 [0.4 to 0.7] | 0.1 [0.0 to 0.1]
  ST6 Month 30: number analyzed (Participants) | 35 | 16
  ST6 Month 30 | 0.2 [0.2 to 0.3] | 0.0 [0.0 to 0.1]

23. Secondary Outcome: GMFR as Compared to Month 18 (Pre-booster) for IgG Against Each OspA Serotype (ST1 to ST6): Booster PP Population
Description: GMFR as compared to Month 18 (pre-booster) for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Month 19, Month 24 and Month 30. The outcome measure was planned to be analyzed for Booster PP population.
Time Frame: Month 18 (from where comparison was done), Month 19, Month 24 and Month 30
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 37 | 18
Fold Rise
  ST1 Month 19 | 51.3 [37.1 to 71.0] | 1.0 [1.0 to 1.0]
  ST1 Month 24: number analyzed (Participants) | 37 | 17
  ST1 Month 24 | 5.5 [4.2 to 7.3] | 0.9 [0.8 to 1.0]
  ST1 Month 30: number analyzed (Participants) | 37 | 17
  ST1 Month 30 | 2.2 [1.7 to 2.8] | 0.9 [0.8 to 1.0]
  ST2 Month 19 | 69.1 [54.2 to 88.0] | 1.0 [0.9 to 1.2]
  ST2 Month 24: number analyzed (Participants) | 37 | 17
  ST2 Month 24 | 8.1 [6.8 to 9.8] | 0.8 [0.6 to 0.9]
  ST2 Month 30: number analyzed (Participants) | 37 | 17
  ST2 Month 30 | 2.8 [2.2 to 3.6] | 0.6 [0.5 to 0.9]
  ST3 Month 19 | 61.7 [46.2 to 82.5] | 0.9 [0.8 to 1.0]
  ST3 Month 24: number analyzed (Participants) | 37 | 17
  ST3 Month 24 | 8.6 [7.0 to 10.4] | 0.8 [0.6 to 1.0]
  ST3 Month 30: number analyzed (Participants) | 37 | 17
  ST3 Month 30 | 3.3 [2.6 to 4.0] | 0.7 [0.5 to 0.9]
  ST4 Month 19 | 57.7 [42.4 to 78.6] | 0.8 [0.7 to 1.0]
  ST4 Month 24: number analyzed (Participants) | 37 | 17
  ST4 Month 24 | 7.0 [5.6 to 8.7] | 0.8 [0.7 to 1.0]
  ST4 Month 30: number analyzed (Participants) | 37 | 17
  ST4 Month 30 | 2.5 [2.0 to 3.2] | 0.7 [0.6 to 0.9]
  ST5 Month 19 | 60.2 [45.1 to 80.4] | 0.8 [0.7 to 1.0]
  ST5 Month 24: number analyzed (Participants) | 37 | 17
  ST5 Month 24 | 6.8 [5.4 to 8.6] | 0.8 [0.7 to 1.0]
  ST5 Month 30: number analyzed (Participants) | 37 | 17
  ST5 Month 30 | 3.0 [2.3 to 3.8] | 0.8 [0.7 to 1.0]
  ST6 Month 19 | 53.5 [39.2 to 73.2] | 1.0 [0.8 to 1.2]
  ST6 Month 24: number analyzed (Participants) | 37 | 17
  ST6 Month 24 | 6.9 [5.4 to 8.9] | 0.9 [0.9 to 1.0]
  ST6 Month 30: number analyzed (Participants) | 37 | 17
  ST6 Month 30 | 2.9 [2.2 to 3.8] | 0.9 [0.7 to 1.0]

24. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Group in Booster PP Population: Group 18 - 49 Years
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24 and Month 30 stratified by age group: 18 - 49 years. The outcome measure was planned to be analyzed for Booster PP population from Day 1 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: as for outcome 19
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 22 | 13
Units per milliliter (U/mL)
  ST1 Day 1 | 20.8 [19.2 to 22.5] | 20.0 [20.0 to 20.0]
  ST1 Day 29 | 21.6 [19.3 to 24.1] | 20.0 [20.0 to 20.0]
  ST1 Day 57 | 22.5 [19.7 to 25.8] | 20.0 [20.0 to 20.0]
  ST1 Day 85: number analyzed (Participants) | 22 | 12
  ST1 Day 85 | 103.1 [60.3 to 176.4] | 62.8 [33.6 to 117.4]
  ST1 Day 180 | 29.2 [23.0 to 37.0] | 21.9 [18.0 to 26.7]
  ST1 Day 208: number analyzed (Participants) | 21 | 12
  ST1 Day 208 | 335.9 [199.7 to 565.0] | 335.3 [189.4 to 593.7]
  ST1 Day 365: number analyzed (Participants) | 22 | 12
  ST1 Day 365 | 39.3 [27.5 to 56.4] | 34.8 [20.6 to 58.7]
  ST1 Day 545 | 24.6 [20.0 to 30.2] | 21.4 [18.4 to 24.9]
  ST1 Month 19 | 1551.7 [943.9 to 2550.8] | 21.4 [18.5 to 24.8]
  ST1 Month 24: number analyzed (Participants) | 22 | 12
  ST1 Month 24 | 142.1 [90.9 to 222.1] | 20.0 [20.0 to 20.0]
  ST1 Month 30: number analyzed (Participants) | 22 | 12
  ST1 Month 30 | 56.4 [37.6 to 84.8] | 20.0 [20.0 to 20.0]
  ST2 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29 | 24.7 [19.3 to 31.7] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 25.7 [18.9 to 35.0] | 20.0 [20.0 to 20.0]
  ST2 Day 85: number analyzed (Participants) | 22 | 12
  ST2 Day 85 | 252.1 [160.9 to 395.1] | 213.1 [110.0 to 412.8]
  ST2 Day 180 | 43.0 [29.5 to 62.6] | 36.4 [22.4 to 59.3]
  ST2 Day 208: number analyzed (Participants) | 21 | 12
  ST2 Day 208 | 608.9 [428.2 to 866.0] | 761.7 [531.8 to 1091.0]
  ST2 Day 365: number analyzed (Participants) | 22 | 12
  ST2 Day 365 | 65.0 [44.5 to 94.8] | 88.8 [53.3 to 148.1]
  ST2 Day 545 | 28.9 [22.6 to 37.0] | 38.3 [26.0 to 56.5]
  ST2 Month 19 | 2199.0 [1423.5 to 3396.9] | 40.2 [28.0 to 57.7]
  ST2 Month 24: number analyzed (Participants) | 22 | 12
  ST2 Month 24 | 230.4 [166.9 to 317.9] | 25.1 [19.3 to 32.7]
  ST2 Month 30: number analyzed (Participants) | 22 | 12
  ST2 Month 30 | 72.8 [45.9 to 115.3] | 20.0 [20.0 to 20.0]
  ST3 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 23.1 [17.1 to 31.1] | 20.0 [20.0 to 20.0]
  ST3 Day 85: number analyzed (Participants) | 22 | 12
  ST3 Day 85 | 280.1 [162.1 to 483.9] | 266.8 [154.9 to 459.4]
  ST3 Day 180 | 52.8 [37.8 to 73.9] | 45.9 [26.6 to 79.4]
  ST3 Day 208: number analyzed (Participants) | 21 | 12
  ST3 Day 208 | 710.0 [476.3 to 1058.3] | 696.6 [449.8 to 1078.7]
  ST3 Day 365: number analyzed (Participants) | 22 | 12
  ST3 Day 365 | 78.1 [53.2 to 114.6] | 91.0 [50.6 to 163.7]
  ST3 Day 545 | 30.4 [22.7 to 40.7] | 41.5 [27.0 to 63.7]
  ST3 Month 19 | 1997.3 [1280.0 to 3116.6] | 37.5 [25.6 to 55.0]
  ST3 Month 24: number analyzed (Participants) | 22 | 12
  ST3 Month 24 | 246.0 [174.9 to 346.2] | 28.3 [20.3 to 39.5]
  ST3 Month 30: number analyzed (Participants) | 22 | 12
  ST3 Month 30 | 96.3 [68.9 to 134.8] | 23.3 [18.5 to 29.2]
  ST4 Day 1 | 21.3 [18.7 to 24.4] | 20.0 [20.0 to 20.0]
  ST4 Day 29 | 22.0 [19.1 to 25.5] | 20.0 [20.0 to 20.0]
  ST4 Day 57 | 23.8 [19.3 to 29.4] | 20.0 [20.0 to 20.0]
  ST4 Day 85: number analyzed (Participants) | 22 | 12
  ST4 Day 85 | 134.8 [82.5 to 220.4] | 105.4 [61.4 to 180.8]
  ST4 Day 180 | 31.1 [23.5 to 41.1] | 29.5 [20.3 to 43.0]
  ST4 Day 208: number analyzed (Participants) | 21 | 12
  ST4 Day 208 | 432.0 [288.2 to 647.4] | 458.6 [306.9 to 685.3]
  ST4 Day 365: number analyzed (Participants) | 22 | 12
  ST4 Day 365 | 45.8 [31.9 to 65.8] | 47.3 [29.9 to 74.9]
  ST4 Day 545 | 29.3 [22.8 to 37.5] | 28.6 [21.4 to 38.2]
  ST4 Month 19 | 1817.7 [1179.3 to 2801.5] | 25.4 [19.3 to 33.4]
  ST4 Month 24: number analyzed (Participants) | 22 | 12
  ST4 Month 24 | 191.7 [138.8 to 264.8] | 22.8 [18.7 to 27.8]
  ST4 Month 30: number analyzed (Participants) | 22 | 12
  ST4 Month 30 | 66.8 [44.8 to 99.5] | 20.0 [20.0 to 20.0]
  ST5 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29 | 21.0 [19.0 to 23.1] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 23.6 [18.1 to 30.6] | 20.0 [20.0 to 20.0]
  ST5 Day 85: number analyzed (Participants) | 22 | 12
  ST5 Day 85 | 120.6 [74.6 to 195.0] | 122.6 [70.7 to 212.7]
  ST5 Day 180 | 27.4 [21.5 to 34.9] | 31.9 [21.4 to 47.4]
  ST5 Day 208: number analyzed (Participants) | 21 | 12
  ST5 Day 208 | 380.7 [238.8 to 607.1] | 506.8 [323.4 to 794.1]
  ST5 Day 365: number analyzed (Participants) | 22 | 12
  ST5 Day 365 | 42.5 [29.7 to 60.9] | 55.0 [32.7 to 92.6]
  ST5 Day 545 | 25.1 [20.5 to 30.7] | 31.6 [21.5 to 46.5]
  ST5 Month 19 | 1600.5 [1002.8 to 2554.6] | 24.4 [18.1 to 32.8]
  ST5 Month 24: number analyzed (Participants) | 22 | 12
  ST5 Month 24 | 160.2 [109.5 to 234.3] | 22.2 [17.6 to 27.9]
  ST5 Month 30: number analyzed (Participants) | 22 | 12
  ST5 Month 30 | 78.1 [57.1 to 106.7] | 22.3 [17.6 to 28.1]
  ST6 Day 1 | 21.5 [18.5 to 24.8] | 20.0 [20.0 to 20.0]
  ST6 Day 29 | 22.7 [18.9 to 27.3] | 20.0 [20.0 to 20.0]
  ST6 Day 57 | 27.3 [20.4 to 36.5] | 20.0 [20.0 to 20.0]
  ST6 Day 85: number analyzed (Participants) | 22 | 12
  ST6 Day 85 | 90.2 [53.9 to 151.0] | 121.4 [72.1 to 204.5]
  ST6 Day 180 | 28.5 [21.7 to 37.5] | 34.4 [21.8 to 54.1]
  ST6 Day 208: number analyzed (Participants) | 21 | 12
  ST6 Day 208 | 346.1 [217.3 to 551.1] | 502.5 [314.1 to 803.8]
  ST6 Day 365: number analyzed (Participants) | 22 | 12
  ST6 Day 365 | 42.8 [28.7 to 63.8] | 63.1 [38.1 to 104.4]
  ST6 Day 545 | 25.4 [20.0 to 32.4] | 28.7 [20.3 to 40.6]
  ST6 Month 19 | 1449.3 [878.4 to 2391.3] | 28.7 [20.3 to 40.6]
  ST6 Month 24: number analyzed (Participants) | 22 | 12
  ST6 Month 24 | 163.8 [115.0 to 233.2] | 25.1 [19.1 to 32.8]
  ST6 Month 30: number analyzed (Participants) | 22 | 12
  ST6 Month 30 | 69.6 [48.1 to 100.7] | 22.1 [17.7 to 27.7]

25. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Group in Booster PP Population: Group 50 - 65 Years
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 1 (Month 0), 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24 and Month 30 stratified by age group: 50 - 65 years. The outcome measure was planned to be analyzed for Booster PP population from Day 1 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: as for outcome 19
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 15 | 5
Units per milliliter (U/mL)
  ST1 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST1 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST1 Day 57 | 22.8 [17.2 to 30.3] | 20.0 [20.0 to 20.0]
  ST1 Day 85 | 53.3 [29.6 to 95.9] | 78.8 [24.0 to 259.4]
  ST1 Day 180 | 25.4 [20.2 to 31.9] | 31.6 [14.3 to 69.6]
  ST1 Day 208: number analyzed (Participants) | 14 | 5
  ST1 Day 208 | 236.6 [124.2 to 450.7] | 386.0 [32.8 to 4546.3]
  ST1 Day 365 | 40.2 [24.4 to 66.0] | 44.1 [4.9 to 396.6]
  ST1 Day 545 | 25.3 [19.0 to 33.8] | 32.3 [8.5 to 122.8]
  ST1 Month 19 | 959.7 [482.2 to 1910.2] | 30.7 [9.4 to 100.7]
  ST1 Month 24 | 130.8 [66.8 to 256.0] | 28.8 [10.5 to 79.3]
  ST1 Month 30 | 50.8 [26.7 to 96.6] | 28.2 [10.8 to 73.5]
  ST2 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29 | 21.4 [18.5 to 24.9] | 20.0 [20.0 to 20.0]
  ST2 Day 57 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 85 | 178.8 [102.1 to 313.1] | 137.8 [33.9 to 559.6]
  ST2 Day 180 | 38.3 [24.2 to 60.5] | 26.8 [11.9 to 60.2]
  ST2 Day 208: number analyzed (Participants) | 14 | 5
  ST2 Day 208 | 602.4 [260.7 to 1391.7] | 557.0 [75.6 to 4104.2]
  ST2 Day 365 | 96.1 [51.6 to 179.2] | 51.1 [7.6 to 344.7]
  ST2 Day 545 | 36.5 [22.5 to 59.2] | 30.4 [9.5 to 96.6]
  ST2 Month 19 | 2187.9 [1198.0 to 3995.8] | 29.3 [10.2 to 84.1]
  ST2 Month 24 | 306.4 [184.2 to 509.5] | 28.4 [10.7 to 75.4]
  ST2 Month 30 | 121.2 [70.6 to 207.9] | 27.3 [11.5 to 64.9]
  ST3 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 57 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 85 | 181.8 [92.4 to 357.8] | 179.8 [57.8 to 559.6]
  ST3 Day 180 | 40.8 [26.0 to 64.1] | 39.0 [11.4 to 133.7]
  ST3 Day 208: number analyzed (Participants) | 14 | 5
  ST3 Day 208 | 530.4 [234.5 to 1199.8] | 599.0 [73.4 to 4891.0]
  ST3 Day 365 | 79.7 [43.1 to 147.3] | 61.6 [6.7 to 566.4]
  ST3 Day 545 | 32.1 [21.6 to 47.6] | 34.9 [7.4 to 163.5]
  ST3 Month 19 | 1803.1 [878.3 to 3701.5] | 31.8 [8.8 to 115.6]
  ST3 Month 24 | 297.8 [183.0 to 484.6] | 30.9 [9.3 to 102.9]
  ST3 Month 30 | 109.9 [66.6 to 181.3] | 29.2 [10.2 to 83.7]
  ST4 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST4 Day 29 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST4 Day 57 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST4 Day 85 | 79.7 [45.8 to 138.7] | 90.2 [28.5 to 285.4]
  ST4 Day 180 | 28.6 [21.4 to 38.4] | 25.8 [12.8 to 52.1]
  ST4 Day 208: number analyzed (Participants) | 14 | 5
  ST4 Day 208 | 306.6 [144.9 to 648.8] | 447.5 [49.6 to 4039.3]
  ST4 Day 365 | 50.0 [30.2 to 82.7] | 44.5 [4.8 to 411.4]
  ST4 Day 545 | 28.1 [20.1 to 39.2] | 39.7 [10.8 to 146.7]
  ST4 Month 19 | 1455.5 [726.5 to 2916.0] | 29.8 [9.9 to 89.8]
  ST4 Month 24 | 214.6 [121.0 to 380.7] | 29.3 [10.2 to 84.1]
  ST4 Month 30 | 81.2 [44.1 to 149.3] | 28.1 [10.9 to 72.0]
  ST5 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST5 Day 29 | 23.8 [17.9 to 31.8] | 20.0 [20.0 to 20.0]
  ST5 Day 57 | 22.8 [18.7 to 27.8] | 20.0 [20.0 to 20.0]
  ST5 Day 85 | 77.7 [44.0 to 137.0] | 139.8 [69.1 to 282.8]
  ST5 Day 180 | 25.4 [19.2 to 33.6] | 33.5 [13.8 to 81.4]
  ST5 Day 208: number analyzed (Participants) | 14 | 5
  ST5 Day 208 | 356.0 [182.9 to 693.0] | 584.1 [104.2 to 3275.4]
  ST5 Day 365 | 45.9 [25.7 to 82.1] | 71.6 [12.7 to 403.9]
  ST5 Day 545 | 24.9 [17.8 to 34.9] | 30.0 [9.8 to 92.1]
  ST5 Month 19 | 1381.6 [772.7 to 2470.1] | 28.5 [10.7 to 75.9]
  ST5 Month 24 | 186.0 [111.8 to 309.2] | 27.6 [11.3 to 67.4]
  ST5 Month 30 | 68.3 [36.3 to 128.6] | 27.0 [11.7 to 62.3]
  ST6 Day 1 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST6 Day 29 | 21.1 [18.8 to 23.6] | 20.0 [20.0 to 20.0]
  ST6 Day 57 | 21.7 [18.3 to 25.7] | 20.0 [20.0 to 20.0]
  ST6 Day 85 | 71.4 [42.1 to 120.9] | 105.4 [27.3 to 407.4]
  ST6 Day 180 | 30.1 [21.4 to 42.4] | 42.2 [17.5 to 102.0]
  ST6 Day 208: number analyzed (Participants) | 14 | 5
  ST6 Day 208 | 360.9 [192.4 to 676.9] | 525.1 [80.5 to 3426.2]
  ST6 Day 365 | 53.4 [28.8 to 98.9] | 78.6 [15.5 to 398.1]
  ST6 Day 545 | 27.6 [19.0 to 40.0] | 30.2 [9.6 to 95.3]
  ST6 Month 19 | 1346.7 [811.0 to 2236.3] | 28.8 [10.5 to 79.3]
  ST6 Month 24 | 210.9 [134.5 to 330.8] | 27.7 [11.2 to 68.5]
  ST6 Month 30 | 86.5 [47.6 to 157.4] | 28.1 [10.9 to 72.5]

26. Secondary Outcome: SCR for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Group in Booster PP Population: Group 18 - 49 Years
Description: SCR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24 and Month 30 stratified by age group: 18 - 49 years was presented in this outcome measure. Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): >=4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants. The outcome measure was planned to be analyzed for Booster PP population from Day 29 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: as for outcome 20
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 22 | 13
Percentage of Participants
  ST1 Day 29 | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 22.8]
  ST1 Day 57 | 9.1 [2.5 to 27.8] | 0.0 [0.0 to 22.8]
  ST1 Day 85: number analyzed (Participants) | 22 | 12
  ST1 Day 85 | 72.7 [51.8 to 86.8] | 66.7 [39.1 to 86.2]
  ST1 Day 180 | 31.8 [16.4 to 52.7] | 7.7 [1.4 to 33.3]
  ST1 Day 208: number analyzed (Participants) | 21 | 12
  ST1 Day 208 | 95.2 [77.3 to 99.2] | 100 [75.8 to 100]
  ST1 Day 365: number analyzed (Participants) | 22 | 12
  ST1 Day 365 | 40.9 [23.3 to 61.3] | 33.3 [13.8 to 60.9]
  ST1 Day 545 | 13.6 [4.7 to 33.3] | 7.7 [1.4 to 33.3]
  ST1 Month 19 | 100 [85.1 to 100] | 7.7 [1.4 to 33.3]
  ST1 Month 24: number analyzed (Participants) | 22 | 12
  ST1 Month 24 | 90.9 [72.2 to 97.5] | 0.0 [0.0 to 24.2]
  ST1 Month 30: number analyzed (Participants) | 22 | 12
  ST1 Month 30 | 63.6 [43.0 to 80.3] | 0.0 [0.0 to 24.2]
  ST2 Day 29 | 13.6 [4.7 to 33.3] | 0.0 [0.0 to 22.8]
  ST2 Day 57 | 13.6 [4.7 to 33.3] | 0.0 [0.0 to 22.8]
  ST2 Day 85: number analyzed (Participants) | 22 | 12
  ST2 Day 85 | 100 [85.1 to 100] | 91.7 [64.6 to 98.5]
  ST2 Day 180 | 50.0 [30.7 to 69.3] | 38.5 [17.7 to 64.5]
  ST2 Day 208: number analyzed (Participants) | 21 | 12
  ST2 Day 208 | 100 [84.5 to 100] | 100 [75.8 to 100]
  ST2 Day 365: number analyzed (Participants) | 22 | 12
  ST2 Day 365 | 72.7 [51.8 to 86.8] | 83.3 [55.2 to 95.3]
  ST2 Day 545 | 31.8 [16.4 to 52.7] | 53.8 [29.1 to 76.8]
  ST2 Month 19 | 100 [85.1 to 100] | 61.5 [35.5 to 82.3]
  ST2 Month 24: number analyzed (Participants) | 22 | 12
  ST2 Month 24 | 100 [85.1 to 100] | 25.0 [8.9 to 53.2]
  ST2 Month 30: number analyzed (Participants) | 22 | 12
  ST2 Month 30 | 63.6 [43.0 to 80.3] | 0.0 [0.0 to 24.2]
  ST3 Day 29 | 0.0 [0.0 to 14.9] | 0.0 [0.0 to 22.8]
  ST3 Day 57 | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 22.8]
  ST3 Day 85: number analyzed (Participants) | 22 | 12
  ST3 Day 85 | 90.9 [72.2 to 97.5] | 100 [75.8 to 100]
  ST3 Day 180 | 68.2 [47.3 to 83.6] | 53.8 [29.1 to 76.8]
  ST3 Day 208: number analyzed (Participants) | 21 | 12
  ST3 Day 208 | 100 [84.5 to 100] | 100 [75.8 to 100]
  ST3 Day 365: number analyzed (Participants) | 22 | 12
  ST3 Day 365 | 77.3 [56.6 to 89.9] | 83.3 [55.2 to 95.3]
  ST3 Day 545 | 31.8 [16.4 to 52.7] | 53.8 [29.1 to 76.8]
  ST3 Month 19 | 100 [85.1 to 100] | 53.8 [29.1 to 76.8]
  ST3 Month 24: number analyzed (Participants) | 22 | 12
  ST3 Month 24 | 100 [85.1 to 100] | 33.3 [13.8 to 60.9]
  ST3 Month 30: number analyzed (Participants) | 22 | 12
  ST3 Month 30 | 90.9 [72.2 to 97.5] | 16.7 [4.7 to 44.8]
  ST4 Day 29 | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 22.8]
  ST4 Day 57 | 9.1 [2.5 to 27.8] | 0.0 [0.0 to 22.8]
  ST4 Day 85: number analyzed (Participants) | 22 | 12
  ST4 Day 85 | 86.4 [66.7 to 95.3] | 91.7 [64.6 to 98.5]
  ST4 Day 180 | 31.8 [16.4 to 52.7] | 30.8 [12.7 to 57.6]
  ST4 Day 208: number analyzed (Participants) | 21 | 12
  ST4 Day 208 | 100 [84.5 to 100] | 100 [75.8 to 100]
  ST4 Day 365: number analyzed (Participants) | 22 | 12
  ST4 Day 365 | 54.5 [34.7 to 73.1] | 66.7 [39.1 to 86.2]
  ST4 Day 545 | 31.8 [16.4 to 52.7] | 38.5 [17.7 to 64.5]
  ST4 Month 19 | 100 [85.1 to 100] | 23.1 [8.2 to 50.3]
  ST4 Month 24: number analyzed (Participants) | 22 | 12
  ST4 Month 24 | 100 [85.1 to 100] | 16.7 [4.7 to 44.8]
  ST4 Month 30: number analyzed (Participants) | 22 | 12
  ST4 Month 30 | 68.2 [47.3 to 83.6] | 0.0 [0.0 to 24.2]
  ST5 Day 29 | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 22.8]
  ST5 Day 57 | 9.1 [2.5 to 27.8] | 0.0 [0.0 to 22.8]
  ST5 Day 85: number analyzed (Participants) | 22 | 12
  ST5 Day 85 | 81.8 [61.5 to 92.7] | 91.7 [64.6 to 98.5]
  ST5 Day 180 | 27.3 [13.2 to 48.2] | 38.5 [17.7 to 64.5]
  ST5 Day 208: number analyzed (Participants) | 21 | 12
  ST5 Day 208 | 95.2 [77.3 to 99.2] | 100 [75.8 to 100]
  ST5 Day 365: number analyzed (Participants) | 22 | 12
  ST5 Day 365 | 50.0 [30.7 to 69.3] | 66.7 [39.1 to 86.2]
  ST5 Day 545 | 22.7 [10.1 to 43.4] | 38.5 [17.7 to 64.5]
  ST5 Month 19 | 100 [85.1 to 100] | 15.4 [4.3 to 42.2]
  ST5 Month 24: number analyzed (Participants) | 22 | 12
  ST5 Month 24 | 95.5 [78.2 to 99.2] | 8.3 [1.5 to 35.4]
  ST5 Month 30: number analyzed (Participants) | 22 | 12
  ST5 Month 30 | 90.9 [72.2 to 97.5] | 8.3 [1.5 to 35.4]
  ST6 Day 29 | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 22.8]
  ST6 Day 57 | 18.2 [7.3 to 38.5] | 0.0 [0.0 to 22.8]
  ST6 Day 85: number analyzed (Participants) | 22 | 12
  ST6 Day 85 | 68.2 [47.3 to 83.6] | 91.7 [64.6 to 98.5]
  ST6 Day 180 | 22.7 [10.1 to 43.4] | 38.5 [17.7 to 64.5]
  ST6 Day 208: number analyzed (Participants) | 21 | 12
  ST6 Day 208 | 95.2 [77.3 to 99.2] | 100 [75.8 to 100]
  ST6 Day 365: number analyzed (Participants) | 22 | 12
  ST6 Day 365 | 40.9 [23.3 to 61.3] | 75.0 [46.8 to 91.1]
  ST6 Day 545 | 13.6 [4.7 to 33.3] | 30.8 [12.7 to 57.6]
  ST6 Month 19 | 100 [85.1 to 100] | 30.8 [12.7 to 57.6]
  ST6 Month 24: number analyzed (Participants) | 22 | 12
  ST6 Month 24 | 95.5 [78.2 to 99.2] | 25.0 [8.9 to 53.2]
  ST6 Month 30: number analyzed (Participants) | 22 | 12
  ST6 Month 30 | 72.7 [51.8 to 86.8] | 8.3 [1.5 to 35.4]

27. Secondary Outcome: SCR for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Group in Booster PP Population: Group 50 - 65 Years
Description: SCR for IgG against each OspA serotype ST1 to ST6, determined by ELISA, at Day 29 (Month 1), 57 (Month 2), 85 (Month 3), 180 (Month 6), 208 (Month 7), 365 (Month 12), 545 (Month 18), Month 19, Month 24, and Month 30 stratified by age group: 50 - 65 years. Seroconversion for ELISA was defined as 1) for participants that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive at a certain time point or 2) for participants that are seropositive at Visit 1 (baseline): >=4-fold rise in IgG antibody titer from Visit 1. SCR was reported as percentage of participants. The outcome measure was planned to be analyzed for Booster PP population from Day 29 to Day 545 of main study phase and from day of vaccination in Month 18 up to Month 30 of booster phase.
Time Frame: as for outcome 20
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 15 | 5
Percentage of Participants
  ST1 Day 29 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST1 Day 57 | 6.7 [1.2 to 29.8] | 0.0 [0.0 to 43.4]
  ST1 Day 85 | 53.3 [30.1 to 75.2] | 80.0 [37.6 to 96.4]
  ST1 Day 180 | 26.7 [10.9 to 52.0] | 40.0 [11.8 to 76.9]
  ST1 Day 208: number analyzed (Participants) | 14 | 5
  ST1 Day 208 | 100 [78.5 to 100] | 100 [56.6 to 100]
  ST1 Day 365 | 46.7 [24.8 to 69.9] | 20.0 [3.6 to 62.4]
  ST1 Day 545 | 20.0 [7.0 to 45.2] | 20.0 [3.6 to 62.4]
  ST1 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST1 Month 24 | 86.7 [62.1 to 96.3] | 20.0 [3.6 to 62.4]
  ST1 Month 30 | 46.7 [24.8 to 69.9] | 20.0 [3.6 to 62.4]
  ST2 Day 29 | 6.7 [1.2 to 29.8] | 0.0 [0.0 to 43.4]
  ST2 Day 57 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST2 Day 85 | 93.3 [70.2 to 98.8] | 80.0 [37.6 to 96.4]
  ST2 Day 180 | 46.7 [24.8 to 69.9] | 20.0 [3.6 to 62.4]
  ST2 Day 208: number analyzed (Participants) | 14 | 5
  ST2 Day 208 | 92.9 [68.5 to 98.7] | 100 [56.6 to 100]
  ST2 Day 365 | 80.0 [54.8 to 93.0] | 40.0 [11.8 to 76.9]
  ST2 Day 545 | 40.0 [19.8 to 64.3] | 20.0 [3.6 to 62.4]
  ST2 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST2 Month 24 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST2 Month 30 | 86.7 [62.1 to 96.3] | 20.0 [3.6 to 62.4]
  ST3 Day 29 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST3 Day 57 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST3 Day 85 | 86.7 [62.1 to 96.3] | 100 [56.6 to 100]
  ST3 Day 180 | 46.7 [24.8 to 69.9] | 40.0 [11.8 to 76.9]
  ST3 Day 208: number analyzed (Participants) | 14 | 5
  ST3 Day 208 | 92.9 [68.5 to 98.7] | 100 [56.6 to 100]
  ST3 Day 365 | 66.7 [41.7 to 84.8] | 40.0 [11.8 to 76.9]
  ST3 Day 545 | 33.3 [15.2 to 58.3] | 20.0 [3.6 to 62.4]
  ST3 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST3 Month 24 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST3 Month 30 | 86.7 [62.1 to 96.3] | 20.0 [3.6 to 62.4]
  ST4 Day 29 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST4 Day 57 | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 43.4]
  ST4 Day 85 | 73.3 [48.0 to 89.1] | 80.0 [37.6 to 96.4]
  ST4 Day 180 | 33.3 [15.2 to 58.3] | 20.0 [3.6 to 62.4]
  ST4 Day 208: number analyzed (Participants) | 14 | 5
  ST4 Day 208 | 92.9 [68.5 to 98.7] | 100 [56.6 to 100]
  ST4 Day 365 | 60.0 [35.7 to 80.2] | 20.0 [3.6 to 62.4]
  ST4 Day 545 | 26.7 [10.9 to 52.0] | 40.0 [11.8 to 76.9]
  ST4 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST4 Month 24 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST4 Month 30 | 80.0 [54.8 to 93.0] | 20.0 [3.6 to 62.4]
  ST5 Day 29 | 13.3 [3.7 to 37.9] | 0.0 [0.0 to 43.4]
  ST5 Day 57 | 13.3 [3.7 to 37.9] | 0.0 [0.0 to 43.4]
  ST5 Day 85 | 73.3 [48.0 to 89.1] | 100 [56.6 to 100]
  ST5 Day 180 | 20.0 [7.0 to 45.2] | 40.0 [11.8 to 76.9]
  ST5 Day 208: number analyzed (Participants) | 14 | 5
  ST5 Day 208 | 100 [78.5 to 100] | 100 [56.6 to 100]
  ST5 Day 365 | 46.7 [24.8 to 69.9] | 80.0 [37.6 to 96.4]
  ST5 Day 545 | 13.3 [3.7 to 37.9] | 20.0 [3.6 to 62.4]
  ST5 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST5 Month 24 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST5 Month 30 | 66.7 [41.7 to 84.8] | 20.0 [3.6 to 62.4]
  ST6 Day 29 | 6.7 [1.2 to 29.8] | 0.0 [0.0 to 43.4]
  ST6 Day 57 | 6.7 [1.2 to 29.8] | 0.0 [0.0 to 43.4]
  ST6 Day 85 | 73.3 [48.0 to 89.1] | 80.0 [37.6 to 96.4]
  ST6 Day 180 | 33.3 [15.2 to 58.3] | 60.0 [23.1 to 88.2]
  ST6 Day 208: number analyzed (Participants) | 14 | 5
  ST6 Day 208 | 100 [78.5 to 100] | 100 [56.6 to 100]
  ST6 Day 365 | 53.3 [30.1 to 75.2] | 80.0 [37.6 to 96.4]
  ST6 Day 545 | 20.0 [7.0 to 45.2] | 20.0 [3.6 to 62.4]
  ST6 Month 19 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST6 Month 24 | 100 [79.6 to 100] | 20.0 [3.6 to 62.4]
  ST6 Month 30 | 73.3 [48.0 to 89.1] | 20.0 [3.6 to 62.4]

28. Secondary Outcome: Percentage of Participants With SAEs During the Entire Booster Phase
Description: as for outcome 11
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 30 (Approximately maximum up to 12 Months)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 7.7 [2.7 to 20.3] | 0.0 [0.0 to 16.8]

29. Secondary Outcome: Percentage of Participants With Related SAEs During the Entire Booster Phase
Description: as for outcome 12
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 30 (Approximately maximum up to 12 Months)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 16.8]

30. Secondary Outcome: Percentage of Participants With Adverse Event of Special Interest (AESIs) During the Entire Booster Phase
Description: as for outcome 13
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 30 (Approximately maximum up to 12 Months)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 2.6 [0.5 to 13.2] | 0.0 [0.0 to 16.8]

31. Secondary Outcome: Percentage of Participants With Related AESIs During the Entire Booster Phase
Description: as for outcome 14
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 30 (Approximately maximum up to 12 Months)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 16.8]

32. Secondary Outcome: Percentage of Participants With Unsolicited AEs During the Booster Phase up to Month 19
Description: An unsolicited AE includes any untoward medical occurrence in a clinical investigation participant temporally associated with the use of investigational product, whether or not related to investigational product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up (more than 6 days after vaccination) for solicited symptoms. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 19 (Approximately for 1 Month)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 15.4 [7.2 to 29.7] | 5.3 [0.9 to 24.6]

33. Secondary Outcome: Percentage of Participants With Related Unsolicited AEs During the Booster Phase up to Month 19
Description: An unsolicited AE included any untoward medical occurrence in a clinical investigation participant temporally associated with the use of investigational product, whether or not related to investigational product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up (more than 6 days after vaccination) for solicited symptoms. Relatedness to study vaccine was assessed by the investigator. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day of vaccination in booster phase (Month 18) up to Month 19 (Approximately for 1 Month)
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants | 5.1 [1.4 to 16.9] | 0.0 [0.0 to 16.8]

34. Secondary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Booster Vaccination
Description: as for outcome 17
Time Frame: Within 7 days after booster vaccination
Population: Booster safety population included all participants who received the booster vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants
  Solicited local AEs | 89.7 [76.4 to 95.9] | 42.1 [23.1 to 63.7]
  Solicited systemic AEs | 51.3 [36.2 to 66.1] | 31.6 [15.4 to 54.0]

35. Secondary Outcome: Percentage of Participants With SAEs, AESIs, Solicited and Unsolicited AEs Stratified by Age Group During the Booster Phase
Description: Percentage of participants with SAEs, AESIs, solicited and unsolicited AEs during booster phase stratified by age group 18-49 years and 50-65 years were reported. SAE: any untoward medical occurrence that at any dose resulted in any of the following outcomes or deemed significant for any other reason: death; required inpatient prolonged existing hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect. AESI: any AEs of scientific/medical concern specific to study vaccine; Solicited AE: predefined reactions at injection site or systemic reactions after each vaccination. Unsolicited AE: any untoward medical occurrence in participant associated with use of study vaccine, whether or not related to study vaccine, reported in addition to solicited and any solicited symptom with onset outside specified period of follow-up.
Time Frame: SAEs and AESIs: From Day of vaccination in booster phase (Month 18) up to Month 30 (Approximately maximum up to 12 Months); AEs: From Day of vaccination in booster phase (Month 18) up to Month 19 (Approximately for 1 Month)
Population: Booster safety population included all participants who received the booster vaccination. Here "Number Analyzed" signifies participants evaluable for this outcome measure at specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
Number analyzed (Participants) | 39 | 19
Percentage of Participants
  SAE: 18-49 Years: number analyzed (Participants) | 22 | 14
  SAE: 18-49 Years | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 21.5]
  SAE: 50-65 Years: number analyzed (Participants) | 17 | 5
  SAE: 50-65 Years | 11.8 [3.3 to 34.3] | 0.0 [0.0 to 43.4]
  AESI: 18-49 Years: number analyzed (Participants) | 22 | 14
  AESI: 18-49 Years | 0.0 [0.0 to 14.9] | 0.0 [0.0 to 21.5]
  AESI: 50-65 Years: number analyzed (Participants) | 17 | 5
  AESI: 50-65 Years | 5.9 [1.0 to 27.0] | 0.0 [0.0 to 43.4]
  Solicited AE: 18-49 Years: number analyzed (Participants) | 22 | 14
  Solicited AE: 18-49 Years | 86.4 [66.7 to 95.3] | 42.9 [21.4 to 67.4]
  Solicited AE: 50-65 Years: number analyzed (Participants) | 17 | 5
  Solicited AE: 50-65 Years | 94.1 [73.0 to 99.0] | 80.0 [37.6 to 96.4]
  Unsolicited AE: 18-49 Years: number analyzed (Participants) | 22 | 14
  Unsolicited AE: 18-49 Years | 9.1 [2.5 to 27.8] | 0.0 [0.0 to 21.5]
  Unsolicited AE: 50-65 Years: number analyzed (Participants) | 17 | 5
  Unsolicited AE: 50-65 Years | 23.5 [9.6 to 47.3] | 20.0 [3.6 to 62.4]

ADVERSE EVENTS:
Time Frame: Solicited AEs (systematic assessment [SA]): up to 7 days after each vaccination; Main study phase: unsolicited AEs (non-SA) including SAEs: up to Day 545; Booster phase: unsolicited AEs (non-SA): From day of vaccination in booster phase (Month 18) up to Month 19 (1 month), SAEs: From day of vaccination in booster phase (Month 18) up to Month 30 (12 months)
Description: Solicited AEs comprised injection site reactions (pain, itching, tenderness, induration [hardening], swelling, erythema [redness]) or systemic reactions (headache, muscle pain, fever [oral], flu-like symptoms, nausea, vomiting, rash, excessive fatigue). Solicited AEs were collected by systematic assessment through participant diaries. Safety population: participants who entered into study and received at least 1 dose of vaccination. For Booster phase, Safety booster population was used.
Groups:
- Main Study Phase: VLA15 With Alum Lower Dose: 0.75 ml injection of VLA15 w/ alum applied at Days 1, 57, and 180. VLA15 is a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate.
- Main Study Phase: VLA15 With Alum Higher Dose: 1 ml injection of VLA15 w/ alum applied at Days 1, 57, and 180. VLA15 is a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate.
- Main Study Phase: Placebo: 1 ml injection of placebo applied at Days 1, 57, and 180. Placebo: phosphate buffered saline (PBS) solution.
Arm/Group | Main Study Phase: VLA15 With Alum Lower Dose | Main Study Phase: VLA15 With Alum Higher Dose | Main Study Phase: Placebo | Booster Phase: VLA15 With Alum Higher Dose | Booster Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/51 | 0/39 | 0/19
Serious Adverse Events (participants affected / at risk) | 4/97 | 4/98 | 2/51 | 3/39 | 0/19
Other Adverse Events (participants affected / at risk) | 94/97 | 97/98 | 40/51 | 35/39 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Phase: VLA15 With Alum Lower Dose (N=97) | Main Study Phase: VLA15 With Alum Higher Dose (N=98) | Main Study Phase: Placebo (N=51) | Booster Phase: VLA15 With Alum Higher Dose (N=39) | Booster Phase: Placebo (N=19)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Phase: VLA15 With Alum Lower Dose (N=97) | Main Study Phase: VLA15 With Alum Higher Dose (N=98) | Main Study Phase: Placebo (N=51) | Booster Phase: VLA15 With Alum Higher Dose (N=39) | Booster Phase: Placebo (N=19)
Injection site pain (General disorders) | 93 | 95 | 16 | 35 | 5 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Injection site erythema (General disorders) | 28 | 41 | 8 | 7 | 3 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Fatigue (General disorders) | 31 | 33 | 13 | 8 | 2 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Injection site induration (General disorders) | 27 | 29 | 1 | 2 | 0 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Injection site swelling (General disorders) | 24 | 32 | 1 | 3 | 1 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Influenza like illness (General disorders) | 18 | 9 | 10 | 1 | 0 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Pyrexia (General disorders) | 8 | 6 | 1 | 0 | 0 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Injection site pruritus (General disorders) | 0 | 5 | 0 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Myalgia (Musculoskeletal and connective tissue disorders) | 54 | 55 | 11 | 11 | 1 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 23 | 8 | 4 | 1 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Headache (Nervous system disorders) | 45 | 45 | 18 | 8 | 4 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Nausea (Gastrointestinal disorders) | 18 | 17 | 6 | 3 | 0 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0 | 1 | 0 — Includes systematic and non-systematic assessments. MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Upper respiratory tract infection (Infections and infestations) | 10 | 7 | 4 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Nasopharyngitis (Infections and infestations) | 7 | 6 | 4 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Sinusitis (Infections and infestations) | 3 | 0 | 5 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Influenza (Infections and infestations) | 2 | 1 | 3 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Red blood cells urine positive (Investigations) | 2 | 2 | 3 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
COVID-19 (Infections and infestations) | 4 | 5 | 1 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 5 | 2 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 — MedDRA v24.0 was used for Main Study Phase (VLA15 lower dose, higher dose and placebo). MedDRA v25.0 was used for Booster Phase (VLA15 higher dose and placebo).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03970733/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03970733/SAP_001.pdf